CLINICAL TRIAL: NCT03765918
Title: A Phase III, Randomized, Open-label Study to Evaluate Pembrolizumab as Neoadjuvant Therapy and in Combination With Standard of Care as Adjuvant Therapy for Stage III-IVA Resectable Locoregionally Advanced Head and Neck Squamous Cell Carcinoma (LA HNSCC)
Brief Title: Study of Pembrolizumab Given Prior to Surgery and in Combination With Radiotherapy Given Post-surgery for Advanced Head and Neck Squamous Cell Carcinoma (MK-3475-689)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-689; MK-3475-689 (Other: MSD); 2022-500254-41-00 (Registry Identifier: EU CT); U1111-1274-2398 (Registry Identifier: UTN); 2017-001139-38 (EudraCT Number)
Record Dates: First submitted 2018-11-06; First posted 2018-12-05 (Actual); Results first posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Head and Neck Neoplasms
Keywords: Programmed Cell Death 1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1 (PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Head and Neck Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab + Standard of Care (SOC) (Experimental): Neoadjuvant treatment: Participants received 200 mg pembrolizumab by intravenous (IV) infusion administered on Day 1 of a 21-day cycle for 2 cycles (up to 6 weeks) prior to surgery.
  Adjuvant treatment: Following surgical resection, participants received 200 mg pembrolizumab, IV infusion, on Day 1 of a 21-day cycle for 15 cycles (up to 45 weeks) plus investigator's choice of SOC treatment regimen consisting of radiotherapy, with or without cisplatin 100 mg/m^2, IV infusion, on Day 1 of a 21-day cycle for 3 cycles (up to 9 weeks).
  Interventions: Biological: Pembrolizumab 200 mg; Radiation: Radiotherapy 60 Gray; Radiation: Radiotherapy 66 Gray; Radiation: Radiotherapy 70 Gray; Drug: Cisplatin 100 mg/m^2
- Standard of Care (SOC) (Active Comparator): Adjuvant treatment: Following surgical resection, participants received investigator's choice of SOC treatment regimen consisting of radiotherapy, with or without cisplatin 100 mg/m^2, IV infusion, on Day 1 of a 21-day cycle for 3 cycles (up to 9 weeks).
  Interventions: Radiation: Radiotherapy 60 Gray; Radiation: Radiotherapy 66 Gray; Radiation: Radiotherapy 70 Gray; Drug: Cisplatin 100 mg/m^2

INTERVENTIONS:
Biological: Pembrolizumab 200 mg — 200 mg administered IV infusion on Day 1 of each 21-day cycle
  Other Names: KEYTRUDA®; MK-3475
  Arms: Pembrolizumab + Standard of Care (SOC)
Radiation: Radiotherapy 60 Gray — Low risk participants administered 2 Gray in 30 fractions. Administered using intensity modulated radiation therapy.
Radiation: Radiotherapy 66 Gray — High risk participants administered 2 Gray in 33 fractions. Administered using intensity modulated radiation therapy.
Radiation: Radiotherapy 70 Gray — Participants with gross residual disease administered 2 Gray in 35 fractions. Administered using intensity modulated radiation therapy.
Drug: Cisplatin 100 mg/m^2 — 100 mg/m^2 administered by IV infusion on Day 1 of each 21-day cycle
  Other Names: Platinol®; Platinol-AQ®

SUMMARY:
This is a randomized, active-controlled, open-label study of pembrolizumab given prior to surgery and pembrolizumab in combination with standard of care radiotherapy (with or without cisplatin), as post-surgical therapy in treatment naïve participants with newly diagnosed Stage III/IVA, resectable, locoregionally advanced, head and neck squamous cell carcinoma (LA-HNSCC). Efficacy outcomes will be stratified by programmed cell death ligand 1 (PD-L1) combined positive score (CPS) status. The primary hypothesis is that pembrolizumab given before surgery and after surgery in combination with radiotherapy (with or without cisplatin) improves event-free survival compared to radiotherapy (with or without cisplatin) given after surgery alone.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically confirmed new diagnosis of resectable, non-metastatic, squamous cell carcinoma that is either: Stage III Human Papillomavirus (HPV) positive oropharyngeal primary that is tumor size (T) 4, lymph node involvement (N) 0-2, no distant metastases (M0); Stage III or IVA oropharyngeal HPV negative; or Stage III or IVA larynx/hypopharynx/oral cavity primaries.
* Is eligible for primary surgery based on investigator decision and per local practice
* Female and male participants of reproductive potential must agree to use adequate contraception throughout the study period and for up to 180 days after the last dose of study therapy.
* Male participants must refrain from donating sperm throughout the study period and for up to 180 days after the last dose of study therapy
* Female participant that is not pregnant or breastfeeding
* Has evaluable tumor burden (measurable and/or non-measurable tumor lesions) assessed by computed tomography (CT) scan or magnetic resonance imaging (MRI), based on Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
* Has provided newly obtained core or excisional biopsy of a tumor lesion not previously irradiated
* Has results from testing of HPV status for oropharyngeal cancer defined as p16
* Has Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 performed within 10 days of randomization

Exclusion Criteria:

* Has Stage T4B and/or N3 locoregionally advanced head and neck squamous cell carcinoma (LA HNSCC) and/or distant metastases
* Has cancer outside of the oropharynx, larynx, and hypopharynx or oral cavity. such as nasopharyngeal, sinus, other para-nasal, or other unknown primary head and neck cancer (HNC)
* Female participant who has a positive urine pregnancy test within 72 hours prior to study start or within 24 hours prior to the start of radiotherapy with or without cisplatin.
* Has received prior therapy with an anti-programmed cell death receptor 1 (PD-1), anti-programmed cell death receptor ligand 1(PD-L1), or anti-programmed cell death receptor ligand 2 (PD-L2) agent or with an agent directed to another co-inhibitory T-cell receptor
* Has received prior radiotherapy treatment or systemic anti-cancer therapy including investigational agents for the HNC under study prior to study start
* Has received a live vaccine within 30 days prior to randomization
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to randomization
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to randomization
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years with the exception of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. in situ cervical cancer or breast carcinoma) that have undergone potentially curative therapy
* Has radiographically detectable (even if asymptomatic and/or previously treated) central nervous system metastases and/or carcinomatous meningitis
* Has Grade ≥2 audiometric hearing loss
* Has Grade ≥2 neuropathy
* Has Grade 3-4 bleeding due to the underlying malignancy
* Has received major surgery or has not recovered adequately from the toxicity and/or complications from the intervention prior to study start
* Has had previous allogeneic tissue/solid organ transplant
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients, radiotherapy, cisplatin or their analogs
* Has an active autoimmune disease that has required systemic treatment in past 2 years
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* Has an active infection requiring systemic therapy
* Has a known history of human immunodeficiency virus (HIV) infection
* Has a known history of or is positive for Hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C (defined as Hepatitis C virus [HCV] ribonucleic acid is detected).
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the investigator
* Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 714 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2026-09-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (192):
- United States (68):
  - Moores Cancer Center ( Site 1885), La Jolla, California
  - University of Southern California Norris Comprehensive Cancer Center ( Site 1850), Los Angeles, California
  - Hoag Memoriall Hospital Presbyterian ( Site 2056), Newport Beach, California
  - UC Davis Health System ( Site 1864), Sacramento, California
  - St. Joseph Heritage Healthcare ( Site 1806), Santa Rosa, California
  - University of Colorado Cancer Center ( Site 1838), Aurora, Colorado
  - MedStar Washington Hospital Center ( Site 2062), Washington D.C., District of Columbia
  - George Washington University Medical Faculty Associates ( Site 2035), Washington D.C., District of Columbia
  - University of Florida ( Site 1832), Gainesville, Florida
  - University of Miami, Sylvester Comprehensive Cancer Center ( Site 2008), Miami, Florida
  - AdventHealth Orlando-AdventHealth Medical Group Hematology & Oncology at Orlando ( Site 2054), Orlando, Florida
  - Orlando Health Cancer Institute ( Site 2061), Orlando, Florida
  - Saint Alphonsus Regional Medical Center ( Site 2021), Boise, Idaho
  - Beacon Cancer Care ( Site 2052), Post Falls, Idaho
  - Rush University Medical Center ( Site 1823), Chicago, Illinois
  - NorthShore University HealthSystem ( Site 1812), Evanston, Illinois
  - Loyola University Medical Center [Maywood, IL] ( Site 1817), Maywood, Illinois
  - University of Kansas Cancer Center ( Site 2004), Westwood, Kansas
  - University of Kentucky Chandler Medical Center-Medical Oncology ( Site 2069), Lexington, Kentucky
  - Ochsner Cancer Institute ( Site 2045), New Orleans, Louisiana
  - University of Maryland ( Site 2031), Baltimore, Maryland
  - Dana Farber Cancer Center ( Site 1873), Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center ( Site 1875), Worcester, Massachusetts
  - Karmanos Cancer Institute ( Site 1870), Detroit, Michigan
  - Henry Ford Health System ( Site 1803), Detroit, Michigan
  - Southdale Cancer Care, University of Minnesota Medical Center- Edina ( Site 2016), Edina, Minnesota
  - University of Missouri Hospital-Otolaryngology - Head and Neck Surgery ( Site 2058), Columbia, Missouri
  - Mercy Clinic Cancer and Hematology - Chub O'Reilly Cancer Center ( Site 1897), Springfield, Missouri
  - Washington University School of Medicine ( Site 1800), St Louis, Missouri
  - St. Vincent Healthcare Frontier Cancer Center ( Site 1818), Billings, Montana
  - Memorial Sloan Kettering Cancer Center Basking Ridge ( Site 2036), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center- Monmouth ( Site 2039), Middletown, New Jersey
  - MSKCC-Bergen ( Site 2037), Montvale, New Jersey
  - Rutgers Cancer Institute of New Jersey ( Site 2071), New Brunswick, New Jersey
  - Rutgers New Jersey Medical School-department of Hematology oncology ( Site 2053), Newark, New Jersey
  - The University of New Mexico Comprehensive Cancer Center ( Site 1882), Albuquerque, New Mexico
  - Erie County Medical Center ( Site 2047), Buffalo, New York
  - Memorial Sloan-Kettering Cancer Center at Commack ( Site 2038), Commack, New York
  - Memorial Sloan-Kettering Cancer Center at West Harrison ( Site 2041), Harrison, New York
  - Monter Cancer Center ( Site 2060), Lake Success, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone Health ( Site 2014), New York, New York
  - Memorial Sloan Kettering Cancer Center ( Site 1857), New York, New York
  - Weill Cornell Medical College ( Site 2050), New York, New York
  - Northwell Health Cancer Institute ( Site 2030), New York, New York
  - Stony Brook University ( Site 2063), Stony Brook, New York
  - Montefiore Einstein Center ( Site 2028), The Bronx, New York
  - Memorial Sloan Kettering Cancer Center - Nassau ( Site 2040), Uniondale, New York
  - Levine Cancer Institute ( Site 2003), Charlotte, North Carolina
  - Wake Forest Compenhensive Cancer Center ( Site 2029), Winston-Salem, North Carolina
  - Sanford Health Roger Maris Cancer Center ( Site 2034), Fargo, North Dakota
  - University Hospitals ( Site 2032), Cleveland, Ohio
  - The Ohio State University ( Site 2012), Columbus, Ohio
  - Providence Portland Medical Center ( Site 1843), Portland, Oregon
  - Kaiser Permanente Center for Health Research-Kaiser Permanente Medical Center ( Site 2022), Portland, Oregon
  - Oregon Health Science University ( Site 1871), Portland, Oregon
  - St. Luke's University Health Network ( Site 1801), Bethlehem, Pennsylvania
  - Sidney Kimmel Cancer Center - Jefferson Health ( Site 2059), Philadelphia, Pennsylvania
  - Allegheny General Hospital ( Site 1833), Pittsburgh, Pennsylvania
  - Sanford Cancer Center Oncology Clinic ( Site 1859), Sioux Falls, South Dakota
  - Avera Cancer Institute- Research ( Site 2070), Sioux Falls, South Dakota
  - Henry Joyce Cancer Clinic ( Site 1827), Nashville, Tennessee
  - UT Southwestern Medical Center ( Site 1841), Dallas, Texas
  - USA Clinical Trials ( Site 2068), San Antonio, Texas
  - University of Utah, Huntsman Cancer Institute ( Site 1855), Salt Lake City, Utah
  - University of Vermont Medical Center ( Site 2009), Burlington, Vermont
  - UVA Health System - Emily Couric Cancer Center ( Site 1826), Charlottesville, Virginia
  - Inova Schar Cancer Institute ( Site 2026), Fairfax, Virginia
  - Seattle Cancer Care Alliance/Univ of Washington Medical Center ( Site 1865), Seattle, Washington
- Argentina (11):
  - Hospital Universitario Austral ( Site 0009), Pilar, Buenos Aires
  - Centro de Educación Médica e Investigaciones Clínicas (CEMIC)-Medical Oncology ( Site 0019), Buenos Aires, Buenos Aires F.D.
  - Hospital Britanico de Buenos Aires ( Site 0012), Ciudad de Buenos Aires, Buenos Aires F.D.
  - Fundacion Estudios Clinicos-Oncology ( Site 0017), Rosario, Santa Fe Province
  - Sanatorio Britanico ( Site 0013), Rosario, Santa Fe Province
  - Instituto de Oncologia de Rosario ( Site 0002), Rosario, Santa Fe Province
  - Hospital Provincial del Centenario ( Site 0008), Rosario, Santa Fe Province
  - IDIM - Instituto de Diagnóstico e Investigaciones Metabólicas ( Site 0016), Buenos Aires
  - Hospital Aleman Buenos Aires Argentina ( Site 0004), Buenos Aires
  - Instituto de Oncología Angel Roffo ( Site 0003), Buenos Aires
  - CER San Juan Centro Polivalente de Asistencia e Investigacion Clinica ( Site 0010), San Juan
- Australia (2):
  - The Crown Princess Mary Cancer Centre - Westmead Hospital ( Site 0051), Westmead, New South Wales
  - Royal Brisbane and Women s Hospital ( Site 0050), Herston, Queensland
- Austria (4):
  - Landeskrankenhaus - Universitatsklinikum Graz ( Site 1902), Graz, Styria
  - Ordensklinikum Linz Gmbh - Barmherzige Schwestern ( Site 1901), Linz, Upper Austria
  - Landeskrankenhaus Salzburg - Universitatklinikum der PMU ( Site 1900), Salzburg
  - Medizinische Universität Wien ( Site 1903), Vienna
- Belgium (3):
  - Hopital de Jolimont ( Site 0103), Haine-Saint-Paul, Hainaut
  - UZ Gent ( Site 0101), Ghent, Oost-Vlaanderen
  - AZ Nikolaas ( Site 0104), Sint-Niklaas, Oost-Vlaanderen
- Brazil (9):
  - Centro Regional Integrado de Oncologia ( Site 0160), Fortaleza, Ceará
  - Hospital Santa Izabel - Santa Casa de Misericordia da Bahia ( Site 0155), Salvador, Estado de Bahia
  - Hospital Marcio Cunha-Unidade de Pesquisa Clínica ( Site 0177), Ipatinga, Minas Gerais
  - Liga Norte Riograndense Contra o Cancer ( Site 0171), Natal, Rio Grande do Norte
  - Hospital Nossa Senhora da Conceicao ( Site 0165), Porto Alegre, Rio Grande do Sul
  - Hospital de Base de Sao Jose de Rio Preto ( Site 0153), São José do Rio Preto, São Paulo
  - Instituto Nacional do Cancer Jose Alencar Gomes da Silva INCA ( Site 0169), Rio de Janeiro
  - Instituto do Cancer do Estado de Sao Paulo - ICESP ( Site 0167), São Paulo
  - BP - A Beneficencia Portuguesa de São Paulo-Medical Oncology ( Site 0175), São Paulo
- Canada (5):
  - Cross Cancer Institute ( Site 0201), Edmonton, Alberta
  - Sunnybrook Research Institute ( Site 0211), Toronto, Ontario
  - Princess Margaret Cancer Centre ( Site 0202), Toronto, Ontario
  - McGill University Health Centre ( Site 0210), Montreal, Quebec
  - CIUSSS de l'Estrie-CHUS ( Site 0209), Sherbrooke, Quebec
- Fundacion Arturo Lopez Perez FALP ( Site 0251), Santiago, Region M. de Santiago, Chile
- Colombia (4):
  - Clinica de la Costa S.A.S. ( Site 0307), Barranquilla, Atlántico
  - Centro de Investigacion Clinica del Country ( Site 0304), Bogotá, Bogota D.C.
  - Oncologos del Occidente S.A. ( Site 0310), Pereira, Risaralda Department
  - Centro Medico Imbanaco de Cali S.A ( Site 0300), Cali, Valle del Cauca Department
- France (7):
  - Centre Antoine Lacassagne ( Site 0351), Nice, Alpes-Maritimes
  - Hopital de la Timone ( Site 0356), Marseille, Bouches-du-Rhone
  - Institut Claudius Regaud IUCT Oncopole ( Site 0355), Toulouse, Haute-Garonne
  - Institut Gustave Roussy ( Site 0353), Villejuif, Val-de-Marne
  - Institut Sainte Catherine ( Site 0352), Avignon, Vaucluse
  - Hopital Europeen Georges Pompidou ( Site 0358), Paris
  - Institut Curie ( Site 0350), Paris
- Germany (12):
  - Universitaetsklinikum Tuebingen - Medizinische Klinik ( Site 0401), Tübingen, Baden-Wurttemberg
  - Universitaetsklinikum Ulm ( Site 0402), Ulm, Baden-Wurttemberg
  - Universitaetsklinikum Erlangen-Strahlenklinik ( Site 0412), Erlangen, Bavaria
  - Klinikum rechts der Isar der Technischen Universitaet ( Site 0409), Munich, Bavaria
  - Klinikum rechts der Isar der Technischen Universität München-HNO Klinik ( Site 0405), München, Bavaria
  - Universitaetsklinikum Frankfurt ( Site 0403), Frankfurt am Main, Hesse
  - Klinikum Kassel GmbH ( Site 0404), Kassel, Hesse
  - Universitaetsklinikum Koeln ( Site 0413), Cologne, North Rhine-Westphalia
  - Universitätsklinikum Schleswig-Holstein ( Site 0411), Lübeck, Schleswig-Holstein
  - SRH Wald-Klinikum Gera GmbH ( Site 0406), Gera, Thuringia
  - Charite Universitätsmedizin Berlin Campus Benjamin Franklin ( Site 0414), Berlin
  - Universitaetsklinikum Hamburg Eppendorf ( Site 0407), Hamburg
- Hungary (4):
  - Pecsi Tudomanyegyetem Onkoterapias Intezet ( Site 0452), Pécs, Baranya
  - Jász-Nagykun-Szolnok Vármegyei Hetényi Géza Kórház ( Site 0450), Szolnok, Jász-Nagykun-Szolnok
  - Eszak-Pesti Centrumkorhaz-Honvedkorhaz ( Site 0453), Budapest
  - Orszagos Onkologiai Intezet ( Site 0454), Budapest
- St. James s Hospital ( Site 0500), Dublin, Ireland
- Israel (5):
  - Rambam Health Care Campus-Oncology Division ( Site 0550), Haifa
  - Hadassah Medical Center. Ein Kerem ( Site 0554), Jerusalem
  - Rabin Medical Center ( Site 0552), Petah Tikva
  - Chaim Sheba Medical Center. ( Site 0553), Ramat Gan
  - Sourasky Medical Center ( Site 0551), Tel Aviv
- Japan (11):
  - Aichi Cancer Center Hospital ( Site 0658), Nagoya, Aichi-ken
  - National Cancer Center Hospital East ( Site 0661), Kashiwa, Chiba
  - Hyogo Cancer Center ( Site 0656), Akashi, Hyōgo
  - Kagawa University Hospital ( Site 0651), Kita-gun, Kagawa-ken
  - Yokohama City University Hospital ( Site 0657), Yokohama, Kanagawa
  - Chiba Cancer Center ( Site 0652), Chiba
  - National Hospital Organization Kyushu Cancer Center ( Site 0660), Fukuoka
  - Hiroshima University Hospital ( Site 0655), Hiroshima
  - National Cancer Center Hospital ( Site 0650), Tokyo
  - Tokyo Medical and Dental University Hospital ( Site 0654), Tokyo
  - Tokyo Medical University Hospital ( Site 0659), Tokyo
- Poland (5):
  - Szpital Specjalistyczny im. Ludwika Rydygiera w Krakowie ( Site 0905), Krakow, Lesser Poland Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy w Warszawie (, Warsaw, Masovian Voivodeship
  - Szpitale Pomorskie Sp. z o.o. ( Site 0935), Gdynia, Pomeranian Voivodeship
  - Narodowy Instytut Onkologii - Oddzial w Gliwicach ( Site 0901), Gliwice, Silesian Voivodeship
  - Wojewodzki Szpital Specjalistyczny im. M. Kopernika w Lodzi ( Site 0920), Lodz, Łódź Voivodeship
- Portugal (4):
  - Hospital de Braga ( Site 0951), Braga
  - CHLN Hospital Santa Maria ( Site 0952), Lisbon
  - Hospital CUF Descobertas ( Site 0953), Lisbon
  - Inst. Portugues de Oncologia de Porto Francisco Gentil EPE ( Site 0950), Porto
- Russia (3):
  - N.N. Blokhin NMRCO ( Site 1005), Moscow, Moscow
  - Republican Clinical Oncology Dispensary of Tatarstan MoH ( Site 1000), Kazan', Tatarstan, Respublika
  - Yaroslavl Regional SBIH Clinical Oncology Hospital ( Site 1001), Yaroslavl, Yaroslavl Oblast
- South Korea (5):
  - Chonnam National University Hwasun Hospital ( Site 0705), Hwasun Gun, Jeonranamdo
  - National Cancer Center ( Site 0702), Goyang-si, Kyonggi-do
  - The Catholic University of Korea St. Vincent s Hospital ( Site 0704), Gyeonggi-do, Kyonggi-do
  - Seoul National University Bundang Hospital ( Site 0703), Seongnam-si, Kyonggi-do
  - Severance Hospital, Yonsei University Health System ( Site 0701), Seoul
- Spain (6):
  - Hospital Germans Trias i Pujol. ICO de Badalona ( Site 1204), Badalona, Barcelona
  - ICO L Hospitalet ( Site 1208), L'Hospitalet de Llobregat, Barcelona
  - Hospital Clinico Universitario de Santiago ( Site 1207), Santiago de Compostela, La Coruna
  - Hospital Vall D Hebron ( Site 1200), Barcelona
  - Hospital Universitario La Paz ( Site 1201), Madrid
  - Hospital Universitario Virgen del Rocio ( Site 1206), Seville
- Switzerland (3):
  - Universitaetsspital Zurich ( Site 1923), Zuerich, Canton of Aargau
  - Istituto Oncologica della Svizzera Italiana (IOSI) ( Site 1921), Bellinzona, Canton Ticino
  - Hopitaux Universitaires de Geneve HUG ( Site 1920), Geneva
- Taiwan (4):
  - Chang Gung Medical Foundation. Kaohsiung Branch ( Site 1303), Kaohsiung City
  - Taichung Veterans General Hospital ( Site 1301), Taichung
  - National Cheng Kung University Hospital ( Site 1302), Tainan
  - National Taiwan University Hospital ( Site 1300), Taipei
- Ukraine (9):
  - Clinical oncology dispensary of Dnipro ( Site 1706), Dnipro, Dnipropetrovsk Oblast
  - Municipal Non-Profit Enterprise City Clinical Hospital 4 of Dnipro City Council ( Site 1705), Dnipro, Dnipropetrovsk Oblast
  - Dnipropetrovsk Regional Hospital n.a. I.I. Mechnikov ( Site 1709), Dnipropetrovsk, Dnipropetrovsk Oblast
  - Ukrainian Center of Tomotherapy ( Site 1708), Kropyvnitskiy, Kirovohrad Oblast
  - PP PPC Acinus Medical and Diagnostic Centre ( Site 1704), Kropyvnytskyi, Kirovohrad Oblast
  - LISOD. Hospital ( Site 1707), Pliuty, Kyiv Oblast
  - Medical Center of Yuriy Spizhenko LLC.-Clinical Trial ( Site 1703), Kapitanivka Village, Kyivska Oblast
  - National Cancer Institute of the MoH of Ukraine ( Site 1702), Kyiv, Kyivska Oblast
  - Kyiv City Clinical Oncology Centre ( Site 1701), Kyiv
- United Kingdom (6):
  - Addenbrooke's Hospital ( Site 1610), Cambridge, Cambridgeshire
  - Castle Hill Hospital ( Site 1601), Cottingham-Hull, Kingston Upon Hull
  - Guy s & St Thomas NHS Foundation Trust ( Site 1604), London, London, City of
  - Royal Marsden Hospital - Fulham Road London ( Site 1609), London, London, City of
  - Imperial Healthcare NHS Trust Charing Cross Hospital ( Site 1603), London, London, City of
  - Weston Park Hospital ( Site 1607), Sheffield

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Uppaluri R, Haddad RI, Tao Y, Le Tourneau C, Lee NY, Westra W, Chernock R, Tahara M, Harrington KJ, Klochikhin AL, Brana I, Vasconcelos Alves G, Hughes BGM, Oliva M, Pinto Figueiredo Lima I, Ueda T, Rutkowski T, Schroeder U, Mauz PS, Fuereder T, Laban S, Oridate N, Popovtzer A, Mach N, Korobko Y, Costa DA, Hooda-Nehra A, Rodriguez CP, Bell RB, Manschot C, Benjamin K, Gumuscu B, Adkins D; KEYNOTE-689 Investigators. Neoadjuvant and Adjuvant Pembrolizumab in Locally Advanced Head and Neck Cancer. N Engl J Med. 2025 Jul 3;393(1):37-50. doi: 10.1056/NEJMoa2415434. Epub 2025 Jun 18. PMID 40532178
- See also: Merck Clinical Trial Information — http://merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26210&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Per protocol, patient-reported outcome (PRO) measures (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 [EORTC QLQ-C30] Global Health Status [GHS]/Quality of Life [QoL][Items 29 and 30], EORTC QLQ-C30 [Items 1-5], EORTC QLQ-Head and Neck Module 35 [H&N35] [Items 35-38], EORTC QLQ-H&N35 [Items 46, 53-54], and EORTC QLQ-H&N35 [Items 31-34] were reported separately for neoadjuvant and adjuvant treatment periods.
Pre-assignment Details: Two participants in the SOC arm received neoadjuvant treatment in error (protocol deviations). One of the participants (who received one cycle of neoadjuvant treatment) was included in the SOC arm for the efficacy and safety analyses per protocol. The other participant (who received 2 cycles of neoadjuvant treatment) was included in the SOC arm for efficacy analysis and in the Pembrolizumab + SOC arm for the safety analysis per protocol.
Period: Overall Study
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Started | 363 | 351
Treated | 360 | 316
Safety Analysis Population (All participants who received ≥1 dose of study treatment: 1 participant in the SOC arm received neoadjuvant treatment, which was a protocol deviation, and this participant was continued in the Pembrolizumab + SOC arm in the study.) | 361 | 315
Efficacy Analysis Population (All randomized participants: 2 participants in the SOC arm received neoadjuvant treatment in error (protocol deviations) and were included in the SOC arm for efficacy analysis.) | 363 | 351
Neoadjuvant Treatment Period: Participants Who Took EORTCQLQ-C30 GHS/QoL (Items 29 & 30) Assessment | 354 | 0
Adjuvant Treatment Period: Participants Who Took EORTCQLQ-C30 GHS/QoL (Items 29 and 30) Assessment | 356 | 306
Neoadjuvant Treatment Period: Participants Who Took EORTCQLQ-C30 (Items 1-5) Assessment | 354 | 0
Adjuvant Treatment Period: Participants Who Took EORTCQLQ-C30 (Items 1-5) Assessment | 356 | 306
Neoadjuvant Treatment Period: Participants Who Took EORTCQLQ-H&N35 (Items 35-38) Assessment | 354 | 0
Adjuvant Treatment Period: Participants Who Took EORTCQLQ-H&N35 (Items 35-38) Assessment | 356 | 306
Neoadjuvant Treatment Period: Participants Who Took EORTCQLQ-H&N35 (Items 46, 53-54) Assessment | 354 | 0
Adjuvant Treatment Period: Participants Who Took EORTCQLQ-H&N35 (Items 46, 53-54) Assessment | 356 | 306
Neoadjuvant Treatment Period: Participants Who Took EORTCQLQ-H&N35 (Items 31-34) Assessment | 354 | 0
Adjuvant Treatment Period: Participants Who Took EORTCQLQ-H&N35 (Items 31-34) Assessment | 356 | 306
Completed | 0 | 0
Not Completed | 363 | 351
Not completed — Death | 109 | 127
Not completed — Lost to Follow-up | 2 | 3
Not completed — Withdrawal by Subject | 12 | 16
Not completed — Participants Ongoing | 240 | 205

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC) | Total
Number analyzed (Participants) | 363 | 351 | 714
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.4 (10.0) | 60.6 (10.0) | 59.9 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 74 | 151
  Male | 286 | 277 | 563
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 55 | 46 | 101
  Not Hispanic or Latino | 300 | 298 | 598
  Unknown or Not Reported | 8 | 7 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 51 | 44 | 95
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 9 | 9 | 18
  White | 284 | 270 | 554
  More than one race | 9 | 20 | 29
  Unknown or Not Reported | 9 | 6 | 15
Primary Tumor Site [Count of Participants; unit: Participants] — The primary tumor site was categorized as tumor in oropharynx, oral cavity, larynx, and hypopharynx. The number of participants with tumor at each site at baseline was presented.
  Participants
    Oropharynx | 35 | 38 | 73
    Oral Cavity | 219 | 213 | 432
    Larynx | 81 | 73 | 154
    Hypopharynx | 28 | 26 | 54
    Missing | 0 | 1 | 1
Overall Cancer Staging at Baseline [Count of Participants; unit: Participants] — American Joint Committee on Cancer 8th edition TNM stratified (PT=primary tumor [size & invasion of nearby tissue], LN=cancerous lymph nodes, Met=distant metastasis). Tumor site stages III: PT (fixated/limited invasion;>2-≥4cm+depth of invasion (DOI) >10mm/>4cm+DOI≥10mm); ipsilateral LN ≤3cm extranodal extension negative(ENE-) (except human papilloma virus [HPV]16+ oropharynx: invasive PT or LN>6cm); IVA: PT (moderate invasion-to adjacent structures[AS]);bilateral/ipsilateral/contralateral LN≤6cm ENE-; IVB: PT (advanced invasion-beyond AS) or LN>6cm ENE±. Higher numbers=more advanced cancer.
  Participants
    III | 90 | 93 | 183
    IVA | 271 | 257 | 528
    IVB | 2 | 0 | 2
    Missing | 0 | 1 | 1
Programmed Cell Death Ligand 1 (PD-L1) Status by Tumor Proportion Score (TPS) [Count of Participants; unit: Participants] — Participants were assessed for their PD-L1 tumor expression level by immunohistochemistry (IHC) assay using tumor tissue from a newly obtained biopsy. The number of participants with TPS <50 and TPS ≥50 at baseline was presented. Higher percentages of PD-L1 TPS staining correspond to higher positivity of PD-L1 on a tumor.
  Participants
    TPS <50% | 257 | 242 | 499
    TPS ≥50% | 103 | 107 | 210
    Missing | 3 | 2 | 5
PD-L1 Status by Combined Positive Score (CPS; CPS10) [Count of Participants; unit: Participants] — The PD-L1 CPS status indicates tumor PD-L1 positivity using both tumor cells and inflammatory cells that are positive for PD-L1 by IHC. The number of participants with CPS <10 and CPS ≥10 at baseline was presented. Participants with a CPS <10 were classified as PD-L1 negative and participants with a CPS ≥10 were classified as PD-L1 positive.
  Participants
    CPS <10 | 126 | 118 | 244
    CPS ≥10 | 234 | 231 | 465
    Missing | 3 | 2 | 5
PD-L1 Status by CPS (CPS1) [Count of Participants; unit: Participants] — The PD-L1 CPS status indicates tumor PD-L1 positivity using both tumor cells and inflammatory cells that are positive for PD-L1 by IHC. The number of participants with CPS <1 and CPS ≥1 at baseline was presented. Participants with a CPS <1 were classified as PD-L1 negative and participants with a CPS ≥1 were classified as PD-L1 positive.
  Participants
    CPS <1 | 13 | 14 | 27
    CPS ≥1 | 347 | 335 | 682
    Missing | 3 | 2 | 5

OUTCOME MEASURES:

1. Secondary Outcome: Major Pathological Response (mPR) Rate
Description: mPR rate was defined as the percentage of participants having ≤10% invasive squamous cell carcinoma within the resected primary tumor specimen and all sampled regional lymph nodes. Per protocol, mPR rate as assessed by blinded independent pathologist review (BIPR) at the time of definitive surgery in all randomized participants was presented.
Time Frame: Up to ~66 months
Population: Efficacy analysis population, which included all randomized participants. Per protocol, two participants in the SOC arm received neoadjuvant treatment in error (protocol deviations) and were included in the SOC arm for efficacy analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 363 | 351
Percentage of Participants | 9.4 [6.6 to 12.8] | 0.0 [0.0 to 1.0]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Other — Difference in percentage (calculated as % Pembrolizumab + SOC arm - % SOC arm) and 95% CI were based on Miettinen & Nurminen method stratified by primary tumor site and tumor stage; p < 0.00001, Stratified Miettinen and Nurminen — One-sided p-value for testing. H0: difference in % = 0 versus H1: difference in % > 0; Difference in Percentage = 9.3, 95% CI 2-sided [6.7 to 12.8]

2. Secondary Outcome: mPR Rate in Participants With PD-L1 CPS ≥10
Description: mPR rate was defined as the percentage of participants having ≤10% invasive squamous cell carcinoma within the resected primary tumor specimen and all sampled regional lymph nodes. Per protocol, mPR rate as assessed by BIPR at the time of definitive surgery in participants with PD-L1 CPS ≥10 was presented.
Time Frame: Up to ~66 months
Population: Efficacy analysis population, which included all randomized participants with PD-L1 CPS ≥10. Per protocol, two participants in the SOC arm received neoadjuvant treatment in error (protocol deviations) and were included in the SOC arm for efficacy analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 234 | 231
Percentage of Participants | 13.7 [9.5 to 18.8] | 0.0 [0.0 to 1.6]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.00001, Stratified Miettinen and Nurminen — One-sided p-value for testing. H0: difference in % = 0 versus H1: difference in % > 0; Difference in Percentage = 13.7, 95% CI 2-sided [9.7 to 18.7]

3. Secondary Outcome: mPR Rate in Participants With PD-L1 CPS ≥1
Description: mPR rate was defined as the percentage of participants having ≤10% invasive squamous cell carcinoma within the resected primary tumor specimen and all sampled regional lymph nodes. Per protocol, mPR rate as assessed by BIPR at the time of definitive surgery in participants with PD-L1 CPS ≥1 was presented.
Time Frame: Up to ~66 months
Population: Efficacy analysis population, which included all randomized participants with PD-L1 CPS ≥1. Per protocol, two participants in the SOC arm received neoadjuvant treatment in error (protocol deviations) and were included in the SOC arm for efficacy analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 347 | 335
Percentage of Participants | 9.8 [6.9 to 13.4] | 0.0 [0.0 to 1.1]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.00001, Stratified Miettinen and Nurminen — One-sided p-value for testing. H0: difference in % = 0 versus H1: difference in % > 0; Difference in Percentage = 9.8, 95% CI 2-sided [7.0 to 13.3]

4. Secondary Outcome: Pathological Complete Response (pCR) Rate
Description: pCR rate was defined as the percentage of participants having no residual invasive squamous cell carcinoma within the resected primary tumor specimen and all sampled regional lymph nodes. The pCR rate as assessed by BIPR at the time of definitive surgery in all randomized participants was presented.
Time Frame: Up to ~66 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 363 | 351
Percentage of Participants | 3.0 [1.5 to 5.4] | 0.0 [0.0 to 1.0]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0006, Stratified Miettinen and Nurminen — One-sided p-value for testing. H0: difference in % = 0 versus H1: difference in % > 0; Difference in Percentage = 3.0, 95% CI 2-sided [1.5 to 5.3]

5. Secondary Outcome: pCR Rate in Participants With PD-L1 CPS ≥10
Description: pCR rate was defined as the percentage of participants having no residual invasive squamous cell carcinoma within the resected primary tumor specimen and all sampled regional lymph nodes. The pCR rate as assessed by BIPR at the time of definitive surgery in all randomized participants with PD-L1 CPS ≥10 was presented.
Time Frame: Up to ~66 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 234 | 231
Percentage of Participants | 4.3 [2.1 to 7.7] | 0.0 [0.0 to 1.6]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0011, Stratified Miettinen and Nurminen — One-sided p-value for testing. H0: difference in % = 0 versus H1: difference in % > 0; Difference in Percentage = 4.2, 95% CI 2-sided [2.1 to 7.6]

6. Secondary Outcome: pCR Rate in Participants With PD-L1 CPS ≥1
Description: pCR rate was defined as the percentage of participants having no residual invasive squamous cell carcinoma within the resected primary tumor specimen and all sampled regional lymph nodes. The pCR rate as assessed by BIPR at the time of definitive surgery in all randomized participants with PD-L1 CPS ≥1 was presented.
Time Frame: Up to ~66 months
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 347 | 335
Percentage of Participants | 3.2 [1.6 to 5.6] | 0.0 [0.0 to 1.1]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0006, Stratified Miettinen and Nurminen — One-sided p-value for testing. H0: difference in % = 0 versus H1: difference in % > 0; Difference in Percentage = 3.1, 95% CI 2-sided [1.6 to 5.6]

7. Secondary Outcome: Neoadjuvant Treatment: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Global Health Status (GHS)/Quality of Life (QoL) (Items 29 & 30) Scale Combined Score at Week 4
Description: EORTC QLQ-C30 is a questionnaire to assess the overall QoL of cancer patients. Participant responses to questions regarding GHS ("How would you rate your overall health during the past week?") and QoL ("How would you rate your overall quality of life during the past week?") were scored on a 7-point scale (1= Very poor to 7=Excellent). The combined score of GHS (Item 29) and QoL (Item 30) were computed by averaging the raw scores of the 2 items and then applying a linear transformation to standardize the average score, so that the combined scores ranged from 0-100. A higher score indicated a better outcome. Per protocol, the change from baseline in GHS and QoL combined score for all randomized participants in the pembrolizumab + SOC arm was presented.
Time Frame: Baseline and Week 4
Population: All randomized participants in the pembrolizumab + SOC treatment group who received at least one dose of study treatment and had at least one EORTC QLQ-C30 assessment data available for this outcome measure at Baseline and at Week 4. Per protocol, this outcome measure was only reported in participants in the pembrolizumab + SOC arm.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 352 | 0
Score on a scale | 2.35 [0.20 to 4.50] |

8. Secondary Outcome: Neoadjuvant Treatment: Change From Baseline in EORTC QLQ-30 GHS/QoL (Items 29 and 30) Scale Combined Score in Participants With PD-L1 CPS ≥10 at Week 4
Description: EORTC QLQ-C30 is a questionnaire to assess the overall QoL of cancer patients. Participant responses to questions regarding GHS ("How would you rate your overall health during the past week?") and QoL ("How would you rate your overall quality of life during the past week?") were scored on a 7-point scale (1= Very poor to 7=Excellent). The combined score of GHS (Item 29) and QoL (Item 30) were computed by averaging the raw scores of the 2 items and then applying a linear transformation to standardize the average score, so that the combined scores ranged from 0-100. A higher score indicated a better outcome. Per protocol, the change from baseline in GHS and QoL combined score for all randomized participants with PD-L1 CPS ≥10 in the pembrolizumab + SOC arm was presented.
Time Frame: Baseline and Week 4
Population: All randomized participants with PD-L1 CPS ≥10 in the pembrolizumab + SOC treatment group who received at least one dose of study treatment and had at least one EORTC QLQ-C30 assessment data available for this outcome measure at Baseline and at Week 4. Per protocol, this outcome measure was only reported in participants in the pembrolizumab + SOC arm.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 225 | 0
Score on a scale | 1.86 [-0.73 to 4.45] |

9. Secondary Outcome: Neoadjuvant Treatment: Change From Baseline in EORTC QLQ-C30 GHS/QOL (Items 29 and 30) Scale Combined Score in Participants With PD-L1 CPS ≥1 at Week 4
Description: EORTC QLQ-C30 is a questionnaire to assess the overall QoL of cancer patients. Participant responses to questions regarding GHS ("How would you rate your overall health during the past week?") and QoL ("How would you rate your overall quality of life during the past week?") were scored on a 7-point scale (1= Very poor to 7=Excellent). The combined score of GHS (Item 29) and QoL (Item 30) were computed by averaging the raw scores of the 2 items and then applying a linear transformation to standardize the average score, so that the combined scores ranged from 0-100. A higher score indicated a better outcome. Per protocol, the change from baseline in GHS and QoL combined score for all randomized participants with PD-L1 CPS ≥1 in the pembrolizumab + SOC arm was presented.
Time Frame: Baseline and Week 4
Population: All randomized participants with PD-L1 CPS ≥1 in the pembrolizumab + SOC treatment group who received at least one dose of study treatment and had at least one EORTC QLQ-C30 assessment data available for this outcome measure at Baseline and at Week 4. Per protocol, this outcome measure was only reported in participants in the pembrolizumab + SOC arm.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 336 | 0
Score on a scale | 2.22 [0.00 to 4.43] |

10. Secondary Outcome: Neoadjuvant Treatment: Change From Baseline in EORTC QLQ-C30 GHS/QoL (Items 29 and 30) Scale Combined Score at Week 6
Description: as for outcome 7
Time Frame: Baseline and Week 6
Population: All randomized participants in the pembrolizumab + SOC treatment group who received at least one dose of study treatment and had at least one EORTC QLQ-C30 assessment data available for this outcome measure at Baseline and at Week 6. Per protocol, this outcome measure was only reported in participants in the pembrolizumab + SOC arm.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 354 | 0
Score on a scale | -0.97 [-3.19 to 1.26] |

11. Secondary Outcome: Neoadjuvant Treatment: Change From Baseline in EORTC QLQ-C30 GHS/QoL (Items 29 and 30) Scale Combined Score in Participants With PD-L1 CPS ≥10 at Week 6
Description: as for outcome 8
Time Frame: Baseline and Week 6
Population: All randomized participants with PD-L1 CPS ≥10 in the pembrolizumab + SOC treatment group who received at least one dose of study treatment and had at least one EORTC QLQ-C30 assessment data available for this outcome measure at Baseline and at Week 6. Per protocol, this outcome measure was only reported in participants in the pembrolizumab + SOC arm.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 227 | 0
Score on a scale | -0.81 [-3.62 to 1.99] |

12. Secondary Outcome: Neoadjuvant Treatment: Change From Baseline in EORTC QLQ-C30 GHS/QoL (Items 29 and 30) Scale Combined Score in Participants With PD-L1 CPS ≥1 at Week 6
Description: as for outcome 9
Time Frame: Baseline and Week 6
Population: All randomized participants with PD-L1 CPS ≥1 in the pembrolizumab + SOC treatment group who received at least one dose of study treatment and had at least one EORTC QLQ-C30 assessment data available for this outcome measure at Baseline and at Week 6. Per protocol, this outcome measure was only reported in participants in the pembrolizumab + SOC arm.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 338 | 0
Score on a scale | -1.22 [-3.52 to 1.08] |

13. Secondary Outcome: Adjuvant Treatment: Change From Baseline in EORTC QLQ-C30 GHS/QoL (Items 29 and 30) Scale Combined Score at Week 25
Description: EORTC QLQ-C30 is a questionnaire to assess the overall QoL of cancer patients. Participant responses to questions regarding GHS ("How would you rate your overall health during the past week?") and QoL ("How would you rate your overall quality of life during the past week?") were scored on a 7-point scale (1= Very poor to 7=Excellent). The combined score of GHS (Item 29) and QoL (Item 30) were computed by averaging the raw scores of the 2 items and then applying a linear transformation to standardize the average score, so that the combined scores ranged from 0-100. A higher score indicated a better outcome. Per protocol, the change from baseline in GHS and QoL combined score for all randomized participants was presented.
Time Frame: Baseline and Week 25
Population: All randomized participants who received at least one dose of study treatment and had at least one EORTC QLQ-C30 assessment data available for this outcome measure at Baseline and at Week 25.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 356 | 306
Score on a scale | 3.69 [1.03 to 6.34] | 4.98 [2.26 to 7.70]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Other — Based on a constrained longitudinal data analysis (cLDA) model with the PRO scores as the response variable with covariates for treatment by study visit interaction, and stratification factors by primary tumor site, tumor stage, and PD-L1 status; p = 0.4671, cLDA model — Two-sided p-value based on cLDA model; Difference in Least Square Means = -1.29, 95% CI 2-sided [-4.78 to 2.20]

14. Secondary Outcome: Adjuvant Treatment: Change From Baseline in EORTC QLQ-C30 GHS/QoL (Items 29 and 30) Scale Combined Score in Participants With PD-L1 CPS ≥10 at Week 25
Description: EORTC QLQ-C30 is a questionnaire to assess the overall QoL of cancer patients. Participant responses to questions regarding GHS ("How would you rate your overall health during the past week?") and QoL ("How would you rate your overall quality of life during the past week?") were scored on a 7-point scale (1= Very poor to 7=Excellent). The combined score of GHS (Item 29) and QoL (Item 30) were computed by averaging the raw scores of the 2 items and then applying a linear transformation to standardize the average score, so that the combined scores ranged from 0-100. A higher score indicated a better outcome. Per protocol, the change from baseline in GHS and QoL combined score for all randomized participants with PD-L1 CPS ≥10 was presented.
Time Frame: Baseline and Week 25
Population: All randomized participants with PD-L1 CPS ≥10 who received at least one dose of study treatment and had at least one EORTC QLQ-C30 assessment data available for this outcome measure at Baseline and at Week 25.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 229 | 203
Score on a scale | 2.13 [-1.15 to 5.40] | 5.16 [1.86 to 8.45]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Other — Based on a cLDA model with the PRO scores as the response variable with covariates for treatment by study visit interaction, and stratification factors by primary tumor site, tumor stage, and PD-L1 status; p = 0.1606, cLDA model — Two-sided p-value based on cLDA model; Difference in Least Square Means = -3.03, 95% CI 2-sided [-7.27 to 1.21]

15. Secondary Outcome: Adjuvant Treatment: Change in EORTC QLQ-C30 GHS/QoL (Items 29 and 30) Scale Combined Score in Participants With PD-L1 CPS ≥1 at Week 25
Description: EORTC QLQ-C30 is a questionnaire to assess the overall QoL of cancer patients. Participant responses to questions regarding GHS ("How would you rate your overall health during the past week?") and QoL ("How would you rate your overall quality of life during the past week?") were scored on a 7-point scale (1= Very poor to 7=Excellent). The combined score of GHS (Item 29) and QoL (Item 30) were computed by averaging the raw scores of the 2 items and then applying a linear transformation to standardize the average score, so that the combined scores ranged from 0-100. A higher score indicated a better outcome. Per protocol, the change from baseline in GHS and QoL combined score for all randomized participants with PD-L1 CPS ≥1 was presented.
Time Frame: Baseline and Week 25
Population: All randomized participants with PD-L1 CPS ≥1 who received at least one dose of study treatment and had at least one EORTC QLQ-C30 assessment data available for this outcome measure at Baseline and at Week 25.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 340 | 291
Score on a scale | 3.62 [0.90 to 6.34] | 5.03 [2.23 to 7.83]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Other — [test comment as in outcome 14, analysis 1]; p = 0.4374, cLDA model — Two-sided p-value based on cLDA model; Difference in Least Square Means = -1.41, 95% CI 2-sided [-4.96 to 2.15]

16. Secondary Outcome: Adjuvant Treatment: Change From Baseline in EORTC QLQ-C30 GHS/QoL (Items 29 and 30) Scale Combined Score at Week 51
Description: as for outcome 13
Time Frame: Baseline and Week 51
Population: All randomized participants who received at least one dose of study treatment and had at least one EORTC QLQ-C30 assessment data available for this outcome measure at Baseline and at Week 51.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 356 | 306
Score on a scale | 4.44 [1.64 to 7.23] | 4.05 [1.13 to 6.97]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Other — [test comment as in outcome 14, analysis 1]; p = 0.8379, cLDA model — Two-sided p-value based on cLDA model; Difference in Least Square Means = 0.39, 95% CI 2-sided [-3.35 to 4.13]

17. Secondary Outcome: Adjuvant Treatment: Change From Baseline in EORTC QLQ-C30 GHS/QoL (Items 29 and 30) Scale Combined Score in Participants With PD-L1 CPS ≥10 at Week 51
Description: as for outcome 14
Time Frame: Baseline and Week 51
Population: All randomized participants with PD-L1 CPS ≥10 who received at least one dose of study treatment and had at least one EORTC QLQ-C30 assessment data available for this outcome measure at Baseline and at Week 51.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 229 | 203
Score on a scale | 4.00 [0.67 to 7.33] | 4.39 [0.90 to 7.87]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Other — [test comment as in outcome 14, analysis 1]; p = 0.8643, cLDA model — Two-sided p-value based on cLDA model; Difference in Least Square Means = -0.39, 95% CI 2-sided [-4.84 to 4.07]

18. Secondary Outcome: Adjuvant Treatment: Change From Baseline in EORTC QLQ-C30 GHS/QoL (Items 29 and 30) Scale Combined Score in Participants With PD-L1 CPS ≥1 at Week 51
Description: as for outcome 15
Time Frame: Baseline and Week 51
Population: All randomized participants with PD-L1 CPS ≥1 who received at least one dose of study treatment and had at least one EORTC QLQ-C30 assessment data available for this outcome measure at Baseline and at Week 51.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 340 | 291
Score on a scale | 4.00 [1.14 to 6.86] | 4.29 [1.29 to 7.29]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Other — [test comment as in outcome 14, analysis 1]; p = 0.8813, cLDA model — Two-sided p-value based on cLDA model; Difference in Least Square Means = -0.29, 95% CI 2-sided [-4.12 to 3.54]

19. Secondary Outcome: Neoadjuvant Treatment: Change From Baseline in Physical Functioning (EORTC QLQ-C30 Items 1-5) Combined Score at Week 4
Description: EORTC QLQ-C30 is a questionnaire to assess the overall QoL of cancer patients. Participant responses to 5 questions about their physical functioning (Items 1 to 5) are scored on a 4-point scale (1=Not at All to 4=Very Much). The combined score of items 1 to 5 was computed by averaging the raw scores of the 5 items and then applying a linear transformation to standardize the average score, so that the combined scores ranged from 0-100. A higher score indicated a better outcome. Per protocol, the change from baseline in EORTC QLQ-C30 physical functioning (Items 1-5) combined score for all randomized participants in the pembrolizumab + SOC arm was presented.
Time Frame: Baseline and Week 4
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 352 | 0
Score on a scale | -2.09 [-3.49 to -0.69] |

20. Secondary Outcome: Neoadjuvant Treatment: Change From Baseline in Physical Functioning (EORTC QLQ-C30 Items 1-5) Combined Score in Participants With PD-L1 CPS ≥10 at Week 4
Description: EORTC QLQ-C30 is a questionnaire to assess the overall QoL of cancer patients. Participant responses to 5 questions about their physical functioning (Items 1 to 5) are scored on a 4-point scale (1=Not at All to 4=Very Much). The combined score of items 1 to 5 was computed by averaging the raw scores of the 5 items and then applying a linear transformation to standardize the average score, so that the combined scores ranged from 0-100. A higher score indicated a better outcome. Per protocol, the change from baseline in EORTC QLQ-C30 physical functioning (Items 1-5) combined score for all randomized participants with PD-L1 CPS ≥10 in the pembrolizumab + SOC arm was presented.
Time Frame: Baseline and Week 4
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 225 | 0
Score on a scale | -2.47 [-4.25 to -0.69] |

21. Secondary Outcome: Neoadjuvant Treatment: Change From Baseline in Physical Functioning (EORTC QLQ-C30 Items 1-5) Combined Score in Participants With PD-L1 CPS ≥1 at Week 4
Description: EORTC QLQ-C30 is a questionnaire to assess the overall QoL of cancer patients. Participant responses to 5 questions about their physical functioning (Items 1 to 5) are scored on a 4-point scale (1=Not at All to 4=Very Much). The combined score of items 1 to 5 was computed by averaging the raw scores of the 5 items and then applying a linear transformation to standardize the average score, so that the combined scores ranged from 0-100. A higher score indicated a better outcome. Per protocol, the change from baseline in EORTC QLQ-C30 physical functioning (Items 1-5) combined score for all randomized participants with PD-L1 CPS ≥1 in the pembrolizumab + SOC arm was presented.
Time Frame: Baseline and Week 4
Population: as for outcome 9
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 336 | 0
Score on a scale | -2.06 [-3.50 to -0.61] |

22. Secondary Outcome: Neoadjuvant Treatment: Change From Baseline in Physical Functioning (EORTC QLQ-C30 Items 1-5) Combined Score at Week 6
Description: as for outcome 19
Time Frame: Baseline and Week 6
Population: as for outcome 10
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 354 | 0
Score on a scale | -3.34 [-4.92 to -1.76] |

23. Secondary Outcome: Neoadjuvant Treatment: Change From Baseline in Physical Functioning (EORTC QLQ-C30 Items 1-5) Combined Score in Participants With PD-L1 CPS ≥10 at Week 6
Description: as for outcome 20
Time Frame: Baseline and Week 6
Population: All randomized participants with PD-L1 CPS ≥10 who received at least one dose of study treatment and had at least one EORTC QLQ-C30 assessment data available for this outcome measure at Baseline and at Week 6. Per protocol, this outcome measure was only reported in participants in the pembrolizumab + SOC arm.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 227 | 0
Score on a scale | -2.42 [-4.53 to -0.32] |

24. Secondary Outcome: Neoadjuvant Treatment: Change From Baseline in Physical Functioning (EORTC QLQ-C30 Items 1-5) Combined Score in Participants With PD-L1 CPS ≥1 at Week 6
Description: as for outcome 21
Time Frame: Baseline and Week 6
Population: All randomized participants with PD-L1 CPS ≥1 who received at least one dose of study treatment and had at least one EORTC QLQ-C30 assessment data available for this outcome measure at Baseline and at Week 6. Per protocol, this outcome measure was only reported in participants in the pembrolizumab + SOC arm.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 338 | 0
Score on a scale | -3.28 [-4.92 to -1.63] |

25. Secondary Outcome: Adjuvant Treatment: Change From Baseline in Physical Functioning (EORTC QLQ-C30 Items 1-5) Combined Score at Week 25
Description: EORTC QLQ-C30 is a questionnaire to assess the overall QoL of cancer patients. Participant responses to 5 questions about their physical functioning (Items 1 to 5) are scored on a 4-point scale (1=Not at All to 4=Very Much). The combined score of items 1 to 5 was computed by averaging the raw scores of the 5 items and then applying a linear transformation to standardize the average score, so that the combined scores ranged from 0-100. A higher score indicated a better outcome. Per protocol, the change from baseline in EORTC QLQ-C30 physical functioning (Items 1-5) combined score for all randomized participants was presented.
Time Frame: Baseline and Week 25
Population: as for outcome 13
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 356 | 306
Score on a scale | -7.48 [-9.72 to -5.25] | -7.83 [-10.15 to -5.50]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Other — [test comment as in outcome 14, analysis 1]; p = 0.8287, cLDA model — Two-sided p-value based on cLDA model; Difference in Least Square Means = 0.34, 95% CI 2-sided [-2.76 to 3.45]

26. Secondary Outcome: Adjuvant Treatment: Change From Baseline in Physical Functioning (EORTC QLQ-C30 Items 1-5) Combined Score in Participants With PD-L1 CPS ≥10 at Week 25
Description: EORTC QLQ-C30 is a questionnaire to assess the overall QoL of cancer patients. Participant responses to 5 questions about their physical functioning (Items 1 to 5) are scored on a 4-point scale (1=Not at All to 4=Very Much). The combined score of items 1 to 5 was computed by averaging the raw scores of the 5 items and then applying a linear transformation to standardize the average score, so that the combined scores ranged from 0-100. A higher score indicated a better outcome. Per protocol, the change from baseline in EORTC QLQ-C30 physical functioning (Items 1-5) combined score for all randomized participants with PD-L1 CPS ≥10 was presented.
Time Frame: Baseline and Week 25
Population: as for outcome 14
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 229 | 203
Score on a scale | -6.22 [-8.91 to -3.53] | -6.75 [-9.47 to -4.03]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Other — [test comment as in outcome 14, analysis 1]; p = 0.7761, cLDA model — Two-sided p-value based on cLDA model; Difference in Least Square Means = 0.53, 95% CI 2-sided [-3.12 to 4.18]

27. Secondary Outcome: Adjuvant Treatment: Change From Baseline in Physical Functioning (EORTC QLQ-C30 Items 1-5) Combined Score in Participants With PD-L1 CPS ≥1 at Week 25
Description: EORTC QLQ-C30 is a questionnaire to assess the overall QoL of cancer patients. Participant responses to 5 questions about their physical functioning (Items 1 to 5) are scored on a 4-point scale (1=Not at All to 4=Very Much). The combined score of items 1 to 5 was computed by averaging the raw scores of the 5 items and then applying a linear transformation to standardize the average score, so that the combined scores ranged from 0-100. A higher score indicated a better outcome. Per protocol, the change from baseline in EORTC QLQ-C30 physical functioning (Items 1-5) combined score for all randomized participants with PD-L1 CPS ≥1 was presented.
Time Frame: Baseline and Week 25
Population: as for outcome 15
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 340 | 291
Score on a scale | -7.42 [-9.71 to -5.13] | -8.07 [-10.46 to -5.68]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Other — [test comment as in outcome 14, analysis 1]; p = 0.6880, cLDA model — Two-sided p-value based on cLDA model; Difference in Least Square Means = 0.65, 95% CI 2-sided [-2.54 to 3.84]

28. Secondary Outcome: Adjuvant Treatment: Change From Baseline in Physical Functioning (EORTC QLQ-C30 Items 1-5) Combined Score at Week 51
Description: as for outcome 25
Time Frame: Baseline and Week 51
Population: as for outcome 16
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 356 | 306
Score on a scale | -6.57 [-8.91 to -4.22] | -5.12 [-7.57 to -2.66]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Other — [test comment as in outcome 14, analysis 1]; p = 0.3858, cLDA model — Two-sided p-value based on cLDA model; Difference in Least Square Means = -1.45, 95% CI 2-sided [-4.73 to 1.83]

29. Secondary Outcome: Adjuvant Treatment: Change From Baseline in Physical Functioning (EORTC QLQ-C30 Items 1-5) Combined Score in Participants With PD-L1 CPS ≥10 at Week 51
Description: as for outcome 26
Time Frame: Baseline and Week 51
Population: as for outcome 17
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 229 | 203
Score on a scale | -7.15 [-10.03 to -4.27] | -4.70 [-7.74 to -1.66]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Other — [test comment as in outcome 14, analysis 1]; p = 0.2370, cLDA model — Two-sided p-value based on cLDA model; Difference in Least Square Means = -2.45, 95% CI 2-sided [-6.53 to 1.62]

30. Secondary Outcome: Adjuvant Treatment: Change From Baseline in Physical Functioning (EORTC QLQ-C30 Items 1-5) Combined Score in Participants With PD-L1 CPS ≥1 at Week 51
Description: as for outcome 27
Time Frame: Baseline and Week 51
Population: as for outcome 18
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 340 | 291
Score on a scale | -6.87 [-9.32 to -4.43] | -5.11 [-7.69 to -2.54]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Other — [test comment as in outcome 14, analysis 1]; p = 0.3138, cLDA model — Two-sided p-value based on cLDA model; Difference in Least Square Means = -1.76, 95% CI 2-sided [-5.20 to 1.67]

31. Secondary Outcome: Neoadjuvant Treatment: Change From Baseline in EORTC QLQ-Head and Neck Module 35 [H&N35] (Items 35-38) Swallowing Combined Score at Week 4
Description: EORTC QLQ-H&N35 is a 35-item questionnaire to assess QoL of head and neck cancer participants and consists of 7 multi-item scales (pain in the mouth, problems with swallowing, senses, speech, social eating, social contact, and sexuality). Participant responses to the swallowing scale (Items 35-38) were scored on a 4-point scale (1=Not at all to 4=Very much). Raw scores were standardized by linear transformation so that scores ranged from 0 to 100; a higher score indicated more problems. Per protocol, the change from baseline in EORTC QLQ-H&N35 swallowing symptoms (Items 35-38) combined score for all randomized participants in the pembrolizumab + SOC arm was presented.
Time Frame: Baseline and Week 4
Population: All randomized participants in the pembrolizumab + SOC treatment group who received at least one dose of study treatment and had at least one EORTC QLQ-H&N35 assessment data available for this outcome measure at Baseline and at Week 4. Per protocol, this outcome measure was only reported in participants in the pembrolizumab + SOC arm.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 352 | 0
Score on a scale | -3.36 [-5.90 to -0.83] |

32. Secondary Outcome: Neoadjuvant Treatment: Change From Baseline in EORTC QLQ-H&N35 (Items 35-38) Swallowing Combined Score in Participants With PD-L1 CPS ≥10 at Week 4
Description: EORTC QLQ-H&N35 is a 35-item questionnaire to assess QoL of head and neck cancer participants and consists of 7 multi-item scales (pain in the mouth, problems with swallowing, senses, speech, social eating, social contact, and sexuality). Participant responses to the swallowing scale (Items 35-38) were scored on a 4-point scale (1=Not at all to 4=Very much). Raw scores were standardized by linear transformation so that scores ranged from 0 to 100; a higher score indicated more problems. Per protocol, the change from baseline in EORTC QLQ-H&N35 swallowing symptoms (Items 35-38) combined score for all randomized participants with PD-L1 CPS ≥10 in the pembrolizumab + SOC arm was presented.
Time Frame: Baseline and Week 4
Population: All randomized participants with PD-L1 CPS ≥10 in the pembrolizumab + SOC treatment group who received at least one dose of study treatment and had at least one EORTC QLQ-H&N35 assessment data available for this outcome measure at Baseline and at Week 4. Per protocol, this outcome measure was only reported in participants in the pembrolizumab + SOC arm.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 225 | 0
Score on a scale | -6.64 [-9.73 to -3.55] |

33. Secondary Outcome: Neoadjuvant Treatment: Change From Baseline in EORTC QLQ-H&N35 (Items 35-38) Swallowing Combined Score in Participants With PD-L1 CPS ≥1 at Week 4
Description: EORTC QLQ-H&N35 is a 35-item questionnaire to assess QoL of head and neck cancer participants and consists of 7 multi-item scales (pain in the mouth, problems with swallowing, senses, speech, social eating, social contact, and sexuality). Participant responses to the swallowing scale (Items 35-38) were scored on a 4-point scale (1=Not at all to 4=Very much). Raw scores were standardized by linear transformation so that scores ranged from 0 to 100; a higher score indicated more problems. Per protocol, the change from baseline in EORTC QLQ-H&N35 swallowing symptoms (Items 35-38) combined score for all randomized participants with PD-L1 CPS ≥1 in the pembrolizumab + SOC arm was presented.
Time Frame: Baseline and Week 4
Population: All randomized participants with PD-L1 CPS ≥1 in the pembrolizumab + SOC treatment group who received at least one dose of study treatment and had at least one EORTC QLQ-H&N35 assessment data available for this outcome measure at Baseline and at Week 4. Per protocol, this outcome measure was only reported in participants in the pembrolizumab + SOC arm.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 336 | 0
Score on a scale | -3.98 [-6.56 to -1.40] |

34. Secondary Outcome: Neoadjuvant Treatment: Change From Baseline in EORTC QLQ-H&N35 (Items 35-38) Swallowing Combined Score at Week 6
Description: as for outcome 31
Time Frame: Baseline and Week 6
Population: All randomized participants in the pembrolizumab + SOC treatment group who received at least one dose of study treatment and had at least one EORTC QLQ-H&N35 assessment data available for this outcome measure at Baseline and at Week 6. Per protocol, this outcome measure was only reported in participants in the pembrolizumab + SOC arm.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 354 | 0
Score on a scale | -2.39 [-4.78 to -0.01] |

35. Secondary Outcome: Neoadjuvant Treatment: Change From Baseline in EORTC QLQ-H&N35 (Items 35-38) Swallowing Combined Score in Participants With PD-L1 CPS ≥10 at Week 6
Description: as for outcome 32
Time Frame: Baseline and Week 6
Population: All randomized participants with PD-L1 CPS ≥10 in the pembrolizumab + SOC treatment group who received at least one dose of study treatment and had at least one EORTC QLQ-H&N35 assessment data available for this outcome measure at Baseline and at Week 6. Per protocol, this outcome measure was only reported in participants in the pembrolizumab + SOC arm.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 227 | 0
Score on a scale | -5.06 [-7.86 to -2.27] |

36. Secondary Outcome: Neoadjuvant Treatment: Change From Baseline in EORTC QLQ-H&N35 (Items 35-38) Swallowing Combined Score in Participants With PD-L1 CPS ≥1 at Week 6
Description: as for outcome 33
Time Frame: Baseline and Week 6
Population: All randomized participants with PD-L1 CPS ≥1 in the pembrolizumab + SOC treatment group who received at least one dose of study treatment and had at least one EORTC QLQ-H&N35 assessment data available for this outcome measure at Baseline and at Week 6. Per protocol, this outcome measure was only reported in participants in the pembrolizumab + SOC arm.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 338 | 0
Score on a scale | -3.05 [-5.47 to -0.63] |

37. Secondary Outcome: Adjuvant Treatment: Change From Baseline in EORTC QLQ-H&N35 (Items 35-38) Swallowing Combined Score at Week 25
Description: EORTC QLQ-H&N35 is a 35-item questionnaire to assess QoL of head and neck cancer participants and consists of 7 multi-item scales (pain in the mouth, problems with swallowing, senses, speech, social eating, social contact, and sexuality). Participant responses to the swallowing scale (Items 35-38) were scored on a 4-point scale (1=Not at all to 4=Very much). Raw scores were standardized by linear transformation so that scores ranged from 0 to 100; a higher score indicated more problems. Per protocol, the change from baseline in EORTC QLQ-H&N35 swallowing symptoms (Items 35-38) combined score for all randomized participants was presented.
Time Frame: Baseline and Week 25
Population: All randomized participants who received at least one dose of study treatment and had at least one EORTC QLQ-H&N35 assessment data available for this outcome measure at Baseline and at Week 25.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 356 | 306
Score on a scale | 4.04 [0.50 to 7.58] | 7.32 [3.69 to 10.95]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Other — [test comment as in outcome 14, analysis 1]; p = 0.1763, cLDA model — Two-sided p-value based on cLDA model; Difference in Least Square Means = -3.28, 95% CI 2-sided [-8.05 to 1.48]

38. Secondary Outcome: Adjuvant Treatment: Change From Baseline in EORTC QLQ-H&N35 (Items 35-38) Swallowing Combined Score in Participants With PD-L1 CPS ≥10 at Week 25
Description: EORTC QLQ-H&N35 is a 35-item questionnaire to assess QoL of head and neck cancer participants and consists of 7 multi-item scales (pain in the mouth, problems with swallowing, senses, speech, social eating, social contact, and sexuality). Participant responses to the swallowing scale (Items 35-38) were scored on a 4-point scale (1=Not at all to 4=Very much). Raw scores were standardized by linear transformation so that scores ranged from 0 to 100; a higher score indicated more problems. Per protocol, the change from baseline in EORTC QLQ-H&N35 swallowing symptoms (Items 35-38) combined score for all randomized participants with PD-L1 CPS ≥10 was presented.
Time Frame: Baseline and Week 25
Population: All randomized participants with PD-L1 CPS ≥10 who received at least one dose of study treatment and had at least one EORTC QLQ-H&N35 assessment data available for this outcome measure at Baseline and at Week 25.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 229 | 203
Score on a scale | 3.89 [-0.47 to 8.24] | 5.06 [0.67 to 9.46]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Other — [test comment as in outcome 14, analysis 1]; p = 0.6882, cLDA model — Two-sided p-value based on cLDA model; Difference in Least Square Means = -1.18, 95% CI 2-sided [-6.95 to 4.59]

39. Secondary Outcome: Adjuvant Treatment: Change From Baseline in EORTC QLQ-H&N35 (Items 35-38) Swallowing Combined Score in Participants With PD-L1 CPS ≥1 at Week 25
Description: EORTC QLQ-H&N35 is a 35-item questionnaire to assess QoL of head and neck cancer participants and consists of 7 multi-item scales (pain in the mouth, problems with swallowing, senses, speech, social eating, social contact, and sexuality). Participant responses to the swallowing scale (Items 35-38) were scored on a 4-point scale (1=Not at all to 4=Very much). Raw scores were standardized by linear transformation so that scores ranged from 0 to 100; a higher score indicated more problems. Per protocol, the change from baseline in EORTC QLQ-H&N35 swallowing symptoms (Items 35-38) combined score for all randomized participants with PD-L1 CPS ≥1 was presented.
Time Frame: Baseline and Week 25
Population: All randomized participants with PD-L1 CPS ≥1 who received at least one dose of study treatment and had at least one EORTC QLQ-H&N35 assessment data available for this outcome measure at Baseline and at Week 25.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 340 | 291
Score on a scale | 4.20 [0.59 to 7.82] | 6.72 [3.00 to 10.45]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Other — [test comment as in outcome 14, analysis 1]; p = 0.3103, cLDA model — Two-sided p-value based on cLDA model; Difference in Least Square Means = -2.52, 95% CI 2-sided [-7.39 to 2.35]

40. Secondary Outcome: Adjuvant Treatment: Change From Baseline in EORTC QLQ-H&N35 (Items 35-38) Swallowing Combined Score at Week 51
Description: as for outcome 37
Time Frame: Baseline and Week 51
Population: All randomized participants who received at least one dose of study treatment and had at least one EORTC QLQ-H&N35 assessment data available for this outcome measure at Baseline and at Week 51.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 356 | 306
Score on a scale | 1.57 [-2.07 to 5.21] | 2.05 [-1.77 to 5.88]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Other — [test comment as in outcome 14, analysis 1]; p = 0.8475, cLDA model — Two-sided p-value based on cLDA model; Difference in Least Square Means = -0.48, 95% CI 2-sided [-5.41 to 4.45]

41. Secondary Outcome: Adjuvant Treatment: Change From Baseline in EORTC QLQ-H&N35 (Items 35-38) Swallowing Combined Score in Participants With PD-L1 CPS ≥10 at Week 51
Description: as for outcome 38
Time Frame: Baseline and Week 51
Population: All randomized participants with PD-L1 CPS ≥10 who received at least one dose of study treatment and had at least one EORTC QLQ-H&N35 assessment data available for this outcome measure at Baseline and at Week 51.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 229 | 203
Score on a scale | 0.50 [-3.90 to 4.90] | 0.93 [-3.74 to 5.59]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Other — [test comment as in outcome 14, analysis 1]; p = 0.8881, cLDA model — Two-sided p-value based on cLDA model; Difference in Least Square Means = -0.42, 95% CI 2-sided [-6.36 to 5.51]

42. Secondary Outcome: Adjuvant Treatment: Change From Baseline in EORTC QLQ-H&N35 (Items 35-38) Swallowing Combined Score in Participants With PD-L1 CPS ≥1 at Week 51
Description: as for outcome 39
Time Frame: Baseline and Week 51
Population: All randomized participants with PD-L1 CPS ≥1 who received at least one dose of study treatment and had at least one EORTC QLQ-H&N35 assessment data available for this outcome measure at Baseline and at Week 51.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 340 | 291
Score on a scale | 1.25 [-2.46 to 4.95] | 1.47 [-2.45 to 5.38]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Other — [test comment as in outcome 14, analysis 1]; p = 0.9307, cLDA model — Two-sided p-value based on cLDA model; Difference in Least Square Means = -0.22, 95% CI 2-sided [-5.22 to 4.78]

43. Secondary Outcome: Neoadjuvant Treatment: Change From Baseline in EORTC QLQ-H&N35 (Items 46, 53-54) Speech Combined Score at Week 4
Description: EORTC QLQ-H&N35 is a 35-item questionnaire to assess QoL of head and neck cancer participants and consists of 7 multi-item scales (pain in the mouth, problems with swallowing, senses, speech, social eating, social contact, and sexuality). Participant responses to the speech scale (Items 46, 53-54) were scored on a 4-point scale (1=Not at all to 4=Very much). Raw scores were standardized by linear transformation so that scores ranged from 0 to 100; a higher score indicated more problems. Per protocol, the change from baseline in EORTC QLQ-H&N35 speech symptoms (Items 46, 53-54) combined score for all randomized participants in the pembrolizumab + SOC arm was presented.
Time Frame: Baseline and Week 4
Population: as for outcome 31
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 352 | 0
Score on a scale | -2.31 [-4.74 to 0.12] |

44. Secondary Outcome: Neoadjuvant Treatment: Change From Baseline in EORTC QLQ-H&N35 (Items 46, 53-54) Speech Combined Score in Participants With PD-L1 CPS ≥10 at Week 4
Description: EORTC QLQ-H&N35 is a 35-item questionnaire to assess QoL of head and neck cancer participants and consists of 7 multi-item scales (pain in the mouth, problems with swallowing, senses, speech, social eating, social contact, and sexuality). Participant responses to the speech scale (Items 46, 53-54) were scored on a 4-point scale (1=Not at all to 4=Very much). Raw scores were standardized by linear transformation so that scores ranged from 0 to 100; a higher score indicated more problems. Per protocol, the change from baseline in EORTC QLQ-H&N35 speech symptoms (Items 46, 53-54) combined score for all randomized participants with PD-L1 CPS ≥10 in the pembrolizumab + SOC arm was presented.
Time Frame: Baseline and Week 4
Population: as for outcome 32
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 225 | 0
Score on a scale | -4.06 [-7.28 to -0.84] |

45. Secondary Outcome: Neoadjuvant Treatment: Change From Baseline in EORTC QLQ-H&N35 (Items 46, 53-54) Speech Combined Score in Participants With PD-L1 CPS ≥1 at Week 4
Description: EORTC QLQ-H&N35 is a 35-item questionnaire to assess QoL of head and neck cancer participants and consists of 7 multi-item scales (pain in the mouth, problems with swallowing, senses, speech, social eating, social contact, and sexuality). Participant responses to the speech scale (Items 46, 53-54) were scored on a 4-point scale (1=Not at all to 4=Very much). Raw scores were standardized by linear transformation so that scores ranged from 0 to 100; a higher score indicated more problems. Per protocol, the change from baseline in EORTC QLQ-H&N35 speech symptoms (Items 46, 53-54) combined score for all randomized participants with PD-L1 CPS ≥1 in the pembrolizumab + SOC arm was presented.
Time Frame: Baseline and Week 4
Population: as for outcome 33
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 336 | 0
Score on a scale | -2.17 [-4.61 to 0.27] |

46. Secondary Outcome: Neoadjuvant Treatment: Change From Baseline in EORTC QLQ-H&N35 (Items 46, 53-54) Speech Combined Score at Week 6
Description: as for outcome 43
Time Frame: Baseline and Week 6
Population: as for outcome 34
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 354 | 0
Score on a scale | -0.74 [-3.14 to 1.67] |

47. Secondary Outcome: Neoadjuvant Treatment: Change From Baseline in EORTC QLQ-H&N35 (Items 46, 53-54) Speech Combined Score in Participants With PD-L1 CPS ≥10 at Week 6
Description: as for outcome 44
Time Frame: Baseline and Week 6
Population: as for outcome 35
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 227 | 0
Score on a scale | -2.84 [-5.96 to 0.27] |

48. Secondary Outcome: Neoadjuvant Treatment: Change From Baseline in EORTC QLQ-H&N35 (Items 46, 53-54) Speech Combined Score in Participants With PD-L1 CPS ≥1 at Week 6
Description: as for outcome 45
Time Frame: Baseline and Week 6
Population: as for outcome 36
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 338 | 0
Score on a scale | -0.76 [-3.22 to 1.70] |

49. Secondary Outcome: Adjuvant Treatment: Change From Baseline in EORTC QLQ-H&N35 (Items 46, 53-54) Speech Combined Score at Week 25
Description: EORTC QLQ-H&N35 is a 35-item questionnaire to assess QoL of head and neck cancer participants and consists of 7 multi-item scales (pain in the mouth, problems with swallowing, senses, speech, social eating, social contact, and sexuality). Participant responses to the speech scale (Items 46, 53-54) were scored on a 4-point scale (1=Not at all to 4=Very much). Raw scores were standardized by linear transformation so that scores ranged from 0 to 100; a higher score indicated more problems. Per protocol, the change from baseline in EORTC QLQ-H&N35 speech symptoms (Items 46, 53-54) combined score for all randomized participants was presented.
Time Frame: Baseline and Week 25
Population: as for outcome 37
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 356 | 306
Score on a scale | 9.80 [6.47 to 13.13] | 8.50 [5.04 to 11.96]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Other — [test comment as in outcome 14, analysis 1]; p = 0.5752, cLDA model — Two-sided p-value based on cLDA model; Difference in Least Square Means = 1.30, 95% CI 2-sided [-3.25 to 5.85]

50. Secondary Outcome: Adjuvant Treatment: Change From Baseline in EORTC QLQ-H&N35 (Items 46, 53-54) Speech Combined Score in Participants With PD-L1 CPS ≥10 at Week 25
Description: EORTC QLQ-H&N35 is a 35-item questionnaire to assess QoL of head and neck cancer participants and consists of 7 multi-item scales (pain in the mouth, problems with swallowing, senses, speech, social eating, social contact, and sexuality). Participant responses to the speech scale (Items 46, 53-54) were scored on a 4-point scale (1=Not at all to 4=Very much). Raw scores were standardized by linear transformation so that scores ranged from 0 to 100; a higher score indicated more problems. Per protocol, the change from baseline in EORTC QLQ-H&N35 speech symptoms (Items 46, 53-54) combined score for all randomized participants with PD-L1 CPS ≥10 was presented.
Time Frame: Baseline and Week 25
Population: as for outcome 38
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 229 | 203
Score on a scale | 8.44 [4.47 to 12.41] | 7.46 [3.36 to 11.57]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Other — [test comment as in outcome 14, analysis 1]; p = 0.7196, cLDA model — Two-sided p-value based on cLDA model; Difference in Least Square Means = 0.98, 95% CI 2-sided [-4.38 to 6.34]

51. Secondary Outcome: Adjuvant Treatment: Change From Baseline in EORTC QLQ-H&N35 (Items 46, 53-54) Speech Combined Score in Participants With PD-L1 CPS ≥1 at Week 25
Description: EORTC QLQ-H&N35 is a 35-item questionnaire to assess QoL of head and neck cancer participants and consists of 7 multi-item scales (pain in the mouth, problems with swallowing, senses, speech, social eating, social contact, and sexuality). Participant responses to the speech scale (Items 46, 53-54) were scored on a 4-point scale (1=Not at all to 4=Very much). Raw scores were standardized by linear transformation so that scores ranged from 0 to 100; a higher score indicated more problems. Per protocol, the change from baseline in EORTC QLQ-H&N35 speech symptoms (Items 46, 53-54) combined score for all randomized participants with PD-L1 CPS ≥1 was presented.
Time Frame: Baseline and Week 25
Population: as for outcome 39
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 340 | 291
Score on a scale | 10.01 [6.64 to 13.39] | 9.27 [5.74 to 12.80]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Other — [test comment as in outcome 14, analysis 1]; p = 0.7522, cLDA model — Two-sided p-value based on cLDA model; Difference in Least Square Means = 0.74, 95% CI 2-sided [-3.88 to 5.37]

52. Secondary Outcome: Adjuvant Treatment: Change From Baseline in EORTC QLQ-H&N35 (Items 46, 53-54) Speech Combined Score at Week 51
Description: as for outcome 49
Time Frame: Baseline and Week 51
Population: as for outcome 40
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 356 | 306
Score on a scale | 5.54 [1.81 to 9.27] | 5.78 [1.91 to 9.65]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Other — [test comment as in outcome 14, analysis 1]; p = 0.9255, cLDA model — Two-sided p-value based on cLDA model; Difference in Least Square Means = -0.24, 95% CI 2-sided [-5.30 to 4.82]

53. Secondary Outcome: Adjuvant Treatment: Change From Baseline in EORTC QLQ-H&N35 (Items 46, 53-54) Speech Combined Score in Participants With PD-L1 CPS ≥10 at Week 51
Description: as for outcome 50
Time Frame: Baseline and Week 51
Population: as for outcome 41
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 229 | 203
Score on a scale | 6.34 [1.65 to 11.03] | 4.11 [-0.81 to 9.04]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Other — [test comment as in outcome 14, analysis 1]; p = 0.4926, cLDA model — Two-sided p-value based on cLDA model; Difference in Least Square Means = 2.22, 95% CI 2-sided [-4.15 to 8.60]

54. Secondary Outcome: Adjuvant Treatment: Change From Baseline in EORTC QLQ-H&N35 (Items 46, 53-54) Speech Combined Score in Participants With PD-L1 CPS ≥1 at Week 51
Description: as for outcome 51
Time Frame: Baseline and Week 51
Population: as for outcome 42
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 340 | 291
Score on a scale | 6.10 [2.27 to 9.92] | 5.10 [1.10 to 9.11]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Other — [test comment as in outcome 14, analysis 1]; p = 0.7087, cLDA model — Two-sided p-value based on cLDA model; Difference in Least Square Means = 0.99, 95% CI 2-sided [-4.23 to 6.21]

55. Secondary Outcome: Neoadjuvant Treatment: Change From Baseline in EORTC QLQ-H&N35 (Items 31-34) Pain Combined Score at Week 4
Description: EORTC QLQ-H&N35 is a 35-item questionnaire to assess QoL of head and neck cancer participants and consists of 7 multi-item scales (pain in the mouth, problems with swallowing, senses, speech, social eating, social contact, and sexuality). Participant responses to the pain scale (Items 31-34) were scored on a 4-point scale (1=Not at all to 4=Very much). Raw scores were standardized by linear transformation so that scores ranged from 0 to 100; a higher score indicated more problems. Per protocol, the change from baseline in EORTC QLQ-H&N35 pain symptoms (Items 31-34) combined score for all randomized participants in the pembrolizumab + SOC arm was presented.
Time Frame: Baseline and Week 4
Population: as for outcome 31
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 352 | 0
Score on a scale | -2.80 [-5.14 to -0.46] |

56. Secondary Outcome: Neoadjuvant Treatment: Change From Baseline in EORTC QLQ-H&N35 (Items 31-34) Pain Combined Score in Participants With PD-L1 CPS ≥10 at Week 4
Description: EORTC QLQ-H&N35 is a 35-item questionnaire to assess QoL of head and neck cancer participants and consists of 7 multi-item scales (pain in the mouth, problems with swallowing, senses, speech, social eating, social contact, and sexuality). Participant responses to the pain scale (Items 31-34) were scored on a 4-point scale (1=Not at all to 4=Very much). Raw scores were standardized by linear transformation so that scores ranged from 0 to 100; a higher score indicated more problems. Per protocol, the change from baseline in EORTC QLQ-H&N35 pain symptoms (Items 31-34) combined score for all randomized participants with PD-L1 CPS ≥10 in the pembrolizumab + SOC arm was presented.
Time Frame: Baseline and Week 4
Population: as for outcome 32
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 225 | 0
Score on a scale | -5.54 [-8.50 to -2.59] |

57. Secondary Outcome: Neoadjuvant Treatment: Change From Baseline in EORTC QLQ-H&N35 (Items 31-34) Pain Combined Score in Participants With PD-L1 CPS ≥1 at Week 4
Description: EORTC QLQ-H&N35 is a 35-item questionnaire to assess QoL of head and neck cancer participants and consists of 7 multi-item scales (pain in the mouth, problems with swallowing, senses, speech, social eating, social contact, and sexuality). Participant responses to the pain scale (Items 31-34) were scored on a 4-point scale (1=Not at all to 4=Very much). Raw scores were standardized by linear transformation so that scores ranged from 0 to 100; a higher score indicated more problems. Per protocol, the change from baseline in EORTC QLQ-H&N35 pain symptoms (Items 31-34) combined score for all randomized participants with PD-L1 CPS ≥1 in the pembrolizumab + SOC arm was presented.
Time Frame: Baseline and Week 4
Population: as for outcome 33
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 336 | 0
Score on a scale | -3.25 [-5.67 to -0.84] |

58. Secondary Outcome: Neoadjuvant Treatment: Change From Baseline in EORTC QLQ-H&N35 (Items 31-34) Pain Combined Score at Week 6
Description: as for outcome 55
Time Frame: Baseline and Week 6
Population: as for outcome 34
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 354 | 0
Score on a scale | -6.27 [-8.68 to -3.87] |

59. Secondary Outcome: Neoadjuvant Treatment: Change From Baseline in EORTC QLQ-H&N35 (Items 31-34) Pain Combined Score in Participants With PD-L1 CPS ≥10 at Week 6
Description: as for outcome 56
Time Frame: Baseline and Week 6
Population: as for outcome 35
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 227 | 0
Score on a scale | -9.14 [-12.17 to -6.11] |

60. Secondary Outcome: Neoadjuvant Treatment: Change From Baseline in EORTC QLQ-H&N35 (Items 31-34) Pain Combined Score in Participants With PD-L1 CPS ≥1 at Week 6
Description: as for outcome 57
Time Frame: Baseline and Week 6
Population: as for outcome 36
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 338 | 0
Score on a scale | -6.76 [-9.23 to -4.28] |

61. Secondary Outcome: Adjuvant Treatment: Change From Baseline in EORTC QLQ-H&N35 (Items 31-34) Pain Combined Score at Week 25
Description: EORTC QLQ-H&N35 is a 35-item questionnaire to assess QoL of head and neck cancer participants and consists of 7 multi-item scales (pain in the mouth, problems with swallowing, senses, speech, social eating, social contact, and sexuality). Participant responses to the pain scale (Items 31-34) were scored on a 4-point scale (1=Not at all to 4=Very much). Raw scores were standardized by linear transformation so that scores ranged from 0 to 100; a higher score indicated more problems. Per protocol, the change from baseline in EORTC QLQ-H&N35 pain symptoms (Items 31-34) combined score for all randomized participants was presented.
Time Frame: Baseline and Week 25
Population: as for outcome 37
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 356 | 306
Score on a scale | -12.16 [-15.20 to -9.12] | -9.41 [-12.52 to -6.29]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Other — [test comment as in outcome 14, analysis 1]; p = 0.1654, cLDA model — Two-sided p-value based on cLDA model; Difference in Least Square Means = -2.75, 95% CI 2-sided [-6.65 to 1.14]

62. Secondary Outcome: Adjuvant Treatment: Change From Baseline in EORTC QLQ-H&N35 (Items 31-34) Pain Combined Score in Participants With PD-L1 CPS ≥10 at Week 25
Description: EORTC QLQ-H&N35 is a 35-item questionnaire to assess QoL of head and neck cancer participants and consists of 7 multi-item scales (pain in the mouth, problems with swallowing, senses, speech, social eating, social contact, and sexuality). Participant responses to the pain scale (Items 31-34) were scored on a 4-point scale (1=Not at all to 4=Very much). Raw scores were standardized by linear transformation so that scores ranged from 0 to 100; a higher score indicated more problems. Per protocol, the change from baseline in EORTC QLQ-H&N35 pain symptoms (Items 31-34) combined score for all randomized participants with PD-L1 CPS ≥10 was presented.
Time Frame: Baseline and Week 25
Population: as for outcome 38
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 229 | 203
Score on a scale | -11.18 [-14.80 to -7.55] | -11.43 [-15.11 to -7.76]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Other — [test comment as in outcome 14, analysis 1]; p = 0.9117, cLDA model — Two-sided p-value based on cLDA model; Difference in Least Square Means = 0.26, 95% CI 2-sided [-4.29 to 4.80]

63. Secondary Outcome: Adjuvant Treatment: Change From Baseline in EORTC QLQ-H&N35 (Items 31-34) Pain Combined Score in Participants With PD-L1 CPS ≥1 at Week 25
Description: EORTC QLQ-H&N35 is a 35-item questionnaire to assess QoL of head and neck cancer participants and consists of 7 multi-item scales (pain in the mouth, problems with swallowing, senses, speech, social eating, social contact, and sexuality). Participant responses to the pain scale (Items 31-34) were scored on a 4-point scale (1=Not at all to 4=Very much). Raw scores were standardized by linear transformation so that scores ranged from 0 to 100; a higher score indicated more problems. Per protocol, the change from baseline in EORTC QLQ-H&N35 pain symptoms (Items 31-34) combined score for all randomized participants with PD-L1 CPS ≥1 was presented.
Time Frame: Baseline and Week 25
Population: as for outcome 39
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 340 | 291
Score on a scale | -11.79 [-14.91 to -8.67] | -9.57 [-12.80 to -6.35]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Other — [test comment as in outcome 14, analysis 1]; p = 0.2808, cLDA model — Two-sided p-value based on cLDA model; Difference in Least Square Means = -2.22, 95% CI 2-sided [-6.25 to 1.82]

64. Secondary Outcome: Adjuvant Treatment: Change From Baseline in EORTC QLQ-H&N35 (Items 31-34) Pain Combined Score at Week 51
Description: as for outcome 61
Time Frame: Baseline and Week 51
Population: as for outcome 40
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 356 | 306
Score on a scale | -14.82 [-17.87 to -11.77] | -12.05 [-15.21 to -8.89]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Other — [test comment as in outcome 14, analysis 1]; p = 0.1577, cLDA model — Two-sided p-value based on cLDA model; Difference in Least Square Means = -2.77, 95% CI 2-sided [-6.62 to 1.08]

65. Secondary Outcome: Adjuvant Treatment: Change From Baseline in EORTC QLQ-H&N35 (Items 31-34) Pain Combined Score in Participants With PD-L1 CPS ≥10 at Week 51
Description: as for outcome 62
Time Frame: Baseline and Week 51
Population: as for outcome 41
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 229 | 203
Score on a scale | -16.34 [-20.12 to -12.56] | -13.53 [-17.47 to -9.60]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Other — [test comment as in outcome 14, analysis 1]; p = 0.2485, cLDA model — Two-sided p-value based on cLDA model; Difference in Least Square Means = -2.81, 95% CI 2-sided [-7.59 to 1.97]

66. Secondary Outcome: Adjuvant Treatment: Change From Baseline in EORTC QLQ-H&N35 (Items 31-34) Pain Combined Score in Participants With PD-L1 CPS ≥1 at Week 51
Description: as for outcome 63
Time Frame: Baseline and Week 51
Population: as for outcome 42
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 340 | 291
Score on a scale | -15.03 [-18.17 to -11.88] | -11.99 [-15.26 to -8.72]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Other — [test comment as in outcome 14, analysis 1]; p = 0.1364, cLDA model — Two-sided p-value based on cLDA model; Difference in Least Square Means = -3.03, 95% CI 2-sided [-7.03 to 0.96]

67. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause. OS for all randomized participants was presented.
Time Frame: Up to ~92 months
Reporting Status: Not Posted

68. Secondary Outcome: OS in Participants With PD-L1 CPS ≥10
Description: OS was defined as the time from randomization to death due to any cause. OS for all randomized participants with PD-L1 CPS ≥10 was presented.
Time Frame: Up to ~92 months
Reporting Status: Not Posted

69. Secondary Outcome: OS in Participants With PD-L1 CPS ≥1
Description: OS was defined as the time from randomization to death due to any cause. OS for all randomized participants with PD-L1 CPS ≥1 was presented.
Time Frame: Up to ~92 months
Reporting Status: Not Posted

70. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE could have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated). The number of participants who experienced one or more AEs was reported.
Time Frame: Up to ~92 months
Reporting Status: Not Posted

71. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE could have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated). The number of participants who discontinued study treatment due to an AE was reported.
Time Frame: Up to ~92 months
Reporting Status: Not Posted

72. Primary Outcome: Event-free Survival (EFS)
Description: EFS was based on Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as assessed by blinded independent central review (BICR) and was defined as the time from randomization to any of the following events: radiographic disease progression (RDP; participants who undergo a definitive biopsy of the progressed lesion and are found to have no histologic evidence of invasive cancer will not meet criteria for an event), RDP during the neoadjuvant phase that precluded surgery, local or distant disease progression or recurrence (as assessed with imaging or biopsy as indicated), or death due to any cause. A secondary malignancy was not considered an EFS event. Per protocol, RECIST 1.1 was modified to allow up to 10 target lesions total (up to 5 per organ). Per protocol, EFS per RECIST 1.1 as assessed by BICR in all randomized participants was presented.
Time Frame: Up to ~66 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 363 | 351
Months | 51.8 [37.5 to NA] — NA = upper limit not reached due to insufficient number of participants with an event. | 30.4 [21.8 to 50.1]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Superiority — Hazard ratio (HR) and associated 95% confidence interval (CI) were based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by primary tumor site and tumor stage; p = 0.00411, Stratified Log Rank; One-sided p-value was based on log-rank test stratified by primary tumor site and tumor stage; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.58 to 0.92]

73. Primary Outcome: EFS in Participants With Programmed Cell Death Ligand 1 (PD-L1) Combined Positive Score (CPS) ≥10
Description: EFS was based on RECIST 1.1 as assessed by BICR and was defined as the time from randomization to any of the following events: RDP (participants who undergo a definitive biopsy of the progressed lesion and are found to have no histologic evidence of invasive cancer will not meet criteria for an event), RDP during the neoadjuvant phase that precluded surgery, local or distant disease progression or recurrence (as assessed with imaging or biopsy as indicated), or death due to any cause. A secondary malignancy was not considered an EFS event. Per protocol, RECIST 1.1 was modified to allow up to 10 target lesions total (up to 5 per organ). Per protocol, EFS per RECIST 1.1 as assessed by BICR in participants with PD-L1 CPS ≥10 was presented.
Time Frame: Up to ~66 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 234 | 231
Months | 59.7 [41.1 to NA] — NA = upper limit not reached due to insufficient number of participants with an event. | 26.9 [18.3 to 51.5]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Superiority — HR and associated 95% CI were based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by primary tumor site and tumor stage; p = 0.00217, Stratified Log Rank; One-sided p-value based on log-rank test stratified by primary tumor site and tumor stage; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.49 to 0.88]

74. Primary Outcome: EFS in Participants With PD-L1 CPS ≥1
Description: EFS was based on RECIST 1.1 as assessed by BICR and was defined as the time from randomization to any of the following events: RDP (participants who undergo a definitive biopsy of the progressed lesion and are found to have no histologic evidence of invasive cancer will not meet criteria for an event), RDP during the neoadjuvant phase that precluded surgery, local or distant disease progression or recurrence (as assessed with imaging or biopsy as indicated), or death due to any cause. A secondary malignancy was not considered an EFS event. Per protocol, RECIST 1.1 was modified to allow up to 10 target lesions total (up to 5 per organ). Per protocol, EFS per RECIST 1.1 as assessed by BICR in participants with PD-L1 CPS ≥1 was presented.
Time Frame: Up to ~66 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 347 | 335
Months | 59.7 [37.9 to NA] — NA = upper limit not reached due to insufficient number of participants with an event. | 29.6 [19.5 to 41.9]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Superiority — [test comment as in outcome 73, analysis 1]; p = 0.00140, Stratified Log Rank; One-sided p-value based on log-rank test stratified by primary tumor site and tumor stage; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.55 to 0.89]

ADVERSE EVENTS:
Time Frame: Up to ~66 months
Description: All-Cause Mortality includes all randomized participants. Serious and Other AEs include the safety analysis population. Per protocol, disease progression of cancer under study was not considered an AE unless considered related to study treatment. Thus, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" & "Disease progression" not related to study treatment are excluded as AEs. Data are reported by treatment received.
Arm/Group | Pembrolizumab + Standard of Care (SOC) | Standard of Care (SOC)
All-Cause Mortality (participants affected / at risk) | 113/363 | 131/351
Serious Adverse Events (participants affected / at risk) | 179/361 | 116/315
Other Adverse Events (participants affected / at risk) | 335/361 | 290/315
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Standard of Care (SOC) (N=361) | Standard of Care (SOC) (N=315)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 5 (5)
Hypercoagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Bradyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiovascular disorder (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Pulmonary valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 4 (4) | 0 (0)
Hypophysitis (Endocrine disorders) | 1 (1) | 0 (0)
Hypopituitarism (Endocrine disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Autoimmune pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 6 (7) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 2 (2)
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 7 (7) | 2 (2)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteric arterial occlusion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 4 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Oesophageal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral cavity fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Salivary gland fistula (Gastrointestinal disorders) | 2 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 6 (6) | 2 (2)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Swollen tongue (Gastrointestinal disorders) | 1 (1) | 0 (0)
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tongue necrosis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2)
Complication associated with device (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 3 (3) | 2 (2)
Face oedema (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 2 (2) | 2 (2)
Impaired healing (General disorders) | 1 (1) | 0 (0)
Implant site thrombosis (General disorders) | 1 (1) | 0 (0)
Inflammation (General disorders) | 1 (1) | 0 (0)
Localised oedema (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 2 (2) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 2 (2)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Procedural failure (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 7 (7) | 1 (1)
Sudden death (General disorders) | 0 (0) | 2 (2)
Swelling face (General disorders) | 1 (2) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 5 (5) | 0 (0)
Anaphylactic shock (Immune system disorders) | 1 (1) | 0 (0)
Transplant rejection (Immune system disorders) | 0 (0) | 1 (1)
Abscess neck (Infections and infestations) | 0 (0) | 1 (1)
Abscess oral (Infections and infestations) | 0 (0) | 1 (1)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 3 (3)
COVID-19 pneumonia (Infections and infestations) | 3 (3) | 2 (2)
Cellulitis (Infections and infestations) | 3 (3) | 1 (1)
Clostridial infection (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 2 (2)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Incision site abscess (Infections and infestations) | 0 (0) | 1 (1)
Infection parasitic (Infections and infestations) | 0 (0) | 1 (1)
Infective glossitis (Infections and infestations) | 1 (1) | 0 (0)
Intervertebral discitis (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella infection (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 2 (2) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Oropharyngeal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 13 (15) | 18 (19)
Pneumonia aspiration (Infections and infestations) | 8 (8) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Postoperative abscess (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 5 (5) | 9 (10)
Pseudomonas infection (Infections and infestations) | 1 (2) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 4 (4) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (2) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 4 (4) | 4 (4)
Sialoadenitis (Infections and infestations) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 5 (6) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1) | 2 (2)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 1 (1)
Submandibular abscess (Infections and infestations) | 1 (1) | 0 (0)
Superinfection (Infections and infestations) | 1 (1) | 0 (0)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 4 (4) | 3 (3)
Wound infection pseudomonas (Infections and infestations) | 0 (0) | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Flap necrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrostomy failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Implant tissue necrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site swelling (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lymphatic duct injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Open fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Osteoradionecrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pharyngeal anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Post procedural complication (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Post procedural fistula (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Postoperative wound complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation skin injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Skin flap necrosis (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tracheal obstruction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 8 (9) | 2 (2)
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1) | 2 (2)
Alcohol intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 2 (2)
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Feeding intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic disorder (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Refeeding syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Bell's palsy (Nervous system disorders) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 2 (2)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 3 (3)
Device dislocation (Product Issues) | 2 (2) | 0 (0)
Device leakage (Product Issues) | 2 (2) | 0 (0)
Internal device exposed (Product Issues) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 6 (6) | 9 (9)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 2 (2)
Immune-mediated nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Prerenal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 2 (2)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Laryngeal fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal fistula (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (6)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 2 (2)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tracheal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticarial dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Arterial haemorrhage (Vascular disorders) | 2 (3) | 1 (1)
Haematoma (Vascular disorders) | 2 (2) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Inferior vena caval occlusion (Vascular disorders) | 0 (0) | 1 (1)
Lymphatic fistula (Vascular disorders) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 2 (2) | 0 (0)
Vascular occlusion (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Standard of Care (SOC) (N=361) | Standard of Care (SOC) (N=315)
Anaemia (Blood and lymphatic system disorders) | 121 (147) | 102 (117)
Tinnitus (Ear and labyrinth disorders) | 20 (23) | 16 (16)
Hyperthyroidism (Endocrine disorders) | 32 (33) | 10 (10)
Hypothyroidism (Endocrine disorders) | 89 (94) | 17 (19)
Constipation (Gastrointestinal disorders) | 96 (115) | 70 (81)
Diarrhoea (Gastrointestinal disorders) | 75 (99) | 31 (34)
Dry mouth (Gastrointestinal disorders) | 81 (87) | 81 (82)
Dyspepsia (Gastrointestinal disorders) | 22 (24) | 10 (10)
Dysphagia (Gastrointestinal disorders) | 99 (108) | 98 (101)
Nausea (Gastrointestinal disorders) | 87 (112) | 84 (106)
Odynophagia (Gastrointestinal disorders) | 31 (34) | 30 (33)
Oral pain (Gastrointestinal disorders) | 48 (56) | 28 (28)
Stomatitis (Gastrointestinal disorders) | 144 (157) | 170 (174)
Vomiting (Gastrointestinal disorders) | 59 (79) | 31 (38)
Asthenia (General disorders) | 39 (46) | 39 (42)
Fatigue (General disorders) | 84 (97) | 52 (53)
Oedema peripheral (General disorders) | 19 (23) | 4 (4)
Pyrexia (General disorders) | 39 (44) | 16 (19)
Oral candidiasis (Infections and infestations) | 36 (45) | 19 (19)
Urinary tract infection (Infections and infestations) | 24 (28) | 8 (8)
Wound infection (Infections and infestations) | 24 (27) | 14 (14)
Procedural pain (Injury, poisoning and procedural complications) | 30 (33) | 32 (32)
Radiation skin injury (Injury, poisoning and procedural complications) | 144 (148) | 150 (151)
Wound dehiscence (Injury, poisoning and procedural complications) | 13 (16) | 20 (23)
Alanine aminotransferase increased (Investigations) | 51 (65) | 29 (37)
Aspartate aminotransferase increased (Investigations) | 42 (51) | 22 (24)
Blood alkaline phosphatase increased (Investigations) | 19 (20) | 9 (9)
Blood creatinine increased (Investigations) | 21 (24) | 21 (24)
Gamma-glutamyltransferase increased (Investigations) | 27 (31) | 7 (8)
Lymphocyte count decreased (Investigations) | 65 (88) | 48 (60)
Neutrophil count decreased (Investigations) | 44 (63) | 61 (87)
Platelet count decreased (Investigations) | 20 (29) | 30 (33)
Weight decreased (Investigations) | 129 (138) | 86 (91)
White blood cell count decreased (Investigations) | 43 (68) | 53 (78)
Decreased appetite (Metabolism and nutrition disorders) | 46 (49) | 41 (43)
Dehydration (Metabolism and nutrition disorders) | 18 (22) | 19 (20)
Hyperglycaemia (Metabolism and nutrition disorders) | 25 (29) | 16 (17)
Hyperkalaemia (Metabolism and nutrition disorders) | 25 (37) | 17 (19)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 35 (44) | 18 (20)
Hypocalcaemia (Metabolism and nutrition disorders) | 22 (23) | 19 (20)
Hypokalaemia (Metabolism and nutrition disorders) | 52 (68) | 39 (49)
Hypomagnesaemia (Metabolism and nutrition disorders) | 34 (48) | 30 (33)
Hyponatraemia (Metabolism and nutrition disorders) | 48 (66) | 24 (32)
Hypophosphataemia (Metabolism and nutrition disorders) | 19 (20) | 17 (17)
Arthralgia (Musculoskeletal and connective tissue disorders) | 31 (39) | 17 (17)
Neck pain (Musculoskeletal and connective tissue disorders) | 32 (35) | 17 (17)
Trismus (Musculoskeletal and connective tissue disorders) | 33 (33) | 22 (23)
Dysarthria (Nervous system disorders) | 16 (16) | 17 (18)
Dysgeusia (Nervous system disorders) | 55 (57) | 60 (60)
Headache (Nervous system disorders) | 30 (38) | 13 (13)
Insomnia (Psychiatric disorders) | 64 (67) | 25 (25)
Cough (Respiratory, thoracic and mediastinal disorders) | 33 (35) | 13 (13)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 (22) | 16 (16)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 24 (26) | 18 (18)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 17 (17) | 19 (19)
Dermatitis (Skin and subcutaneous tissue disorders) | 22 (23) | 21 (21)
Erythema (Skin and subcutaneous tissue disorders) | 13 (15) | 19 (19)
Pruritus (Skin and subcutaneous tissue disorders) | 38 (41) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 40 (53) | 5 (5)
Hypertension (Vascular disorders) | 27 (30) | 14 (20)
Lymphoedema (Vascular disorders) | 26 (27) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. In this case, a coordinating investigator will be designated by mutual agreement. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-29): https://cdn.clinicaltrials.gov/large-docs/18/NCT03765918/Prot_SAP_000.pdf